# **Clinical Study Protocol**



## INCB 18424-271 / NCT02953678

## A Single-Cohort, Phase 2 Study of Ruxolitinib in Combination With Corticosteroids for the Treatment of Steroid-Refractory Acute Graft-Versus-Host Disease

| Product: | INCB018424 |
|---|---|
| IND Number: | 77456 |
| Phase of Study: | 2 |
| Sponsor: | Incyte Corporation<br>1801 Augustine Cut-Off<br>Wilmington, DE 19803 |
| Date of Protocol: | 14 JUN 2016 |
| Date of Amendment 1: | 12 SEP 2016 |
| Date of Amendment 2: | 04 OCT 2016 |

This study will be performed in accordance with ethical principles that have their origin in the Declaration of Helsinki and conducted in adherence to the study Protocol, Good Clinical Practices as defined in Title 21 of the US Code of Federal Regulations Parts 11, 50, 54, 56, and 312 as well as ICH GCP consolidated guidelines (E6) and applicable regulatory requirements.

The information in this document is confidential. No part of this information may be duplicated, referenced, or transmitted in any form or by any means (electronic, mechanical, photocopy, recording, or otherwise) without the prior written consent of Incyte Corporation.

(Signature of Investigator)

## INVESTIGATOR'S AGREEMENT

| ved |
|-----|

(Date)

## **SYNOPSIS**

| b | STNOPSIS | |
|---|---|---|
| N | Name of Investigational Product: INCB018424 | |
| | <b>Title of Study:</b> A Single-Cohort, Phase 2 Study of Ruxolitinib in Combination With Corticosteroids for the Treatment of Steroid-Refractory Acute Graft-Versus-Host Disease | |
| P | Protocol Number: INCB 18424-271 Study Phase: 2 | |
| C | bjectives and Endpoints: | |
| | Primary Objective | Primary Endpoint |
| | Assess the efficacy of ruxolitinib in combination with corticosteroids in subjects with Grade II to IV steroid-refractory acute graft-versus-host disease (GVHD). | Overall response rate (ORR) at Day 28, defined as the proportion of subjects demonstrating a complete response (CR), very good partial response (VGPR), or partial response (PR). |
| | Secondary Objectives | Secondary Endpoints |
| | Assess additional response and longer-term efficacy outcomes in the study population. | Key secondary endpoint: Six-month duration of response (DOR), defined as the time from first response until GVHD progression or death. DOR will be assessed when all subjects complete the Day 180 visit. ORR, defined as the proportion of subjects demonstrating |
| | | a CR, VGPR, PR at Days 14, 56, and 100. Three-month DOR, defined as the time from first response until GVHD progression or death, when all subjects complete the Day 84 visit. Nonrelapse mortality (NRM), defined as the proportion of subjects who died due to causes other than malignancy relapse at Months 6, 9, 12, and 24. |
| | | Relapse rate, defined as the proportion of subjects whose underlying malignancy relapses. |
| | | Relapse-related mortality rate, defined as the proportion of subjects whose malignancy relapses and has a fatal outcome. |
| | | Failure-free survival (FFS), defined as the proportion of subjects who are still alive, have not relapsed, have not required additional therapy for acute GVHD, and have not demonstrated signs or symptoms of chronic GVHD, at Month 6. |
| | | Overall survival (OS), defined as the time from study enrollment to death due to any cause. |
| | Assess the incidence and severity of adverse events (AEs) and serious adverse events (SAEs). | Summaries of clinical safety data (eg, AEs, infections) will be tabulated and listed. |
| | Evaluate the pharmacokinetics of ruxolitinib when administered in combination with corticosteroids. | Maximum observed plasma drug concentration $(C_{max})$ , minimum observed plasma drug concentration $(C_{min})$ , time of maximum observed plasma drug concentration $(t_{max})$ , area under the plasma drug concentration versus time curve (AUC), and apparent clearance of study drug from plasma (CL/F). |



#### **Overall Study Design:**

This is an open-label, single-cohort, multicenter Phase 2 study of ruxolitinib in combination with corticosteroids for the treatment of steroid-refractory Grades II to IV acute GVHD. Eligible subjects will begin treatment at 5 mg twice daily (BID) ruxolitinib; if hematologic parameters are stable and no treatment-related toxicity is observed after the first 3 days of treatment, the dose may be increased to 10 mg BID. Ruxolitinib may be tapered after Day 180 provided the subject has achieved CR or VGPR and corticosteroids have been discontinued for at least 8 weeks. Corticosteroids will be administered at a starting dose of 2.0 mg/kg per day (unless otherwise indicated) on Day 1 and will be tapered as appropriate. Subjects will receive study treatment until treatment failure (progression of GVHD, no response, or requiring additional systemic therapy), unacceptable toxicity, or death. Continued use of anti-infective medications, GVHD prophylaxis medications (including calcineurin inhibitors), transfusion support, and topical steroid therapy is permitted.

Severity of GVHD will be assessed from screening through end of treatment (EOT) using the Mount Sinai Acute GVHD International Consortium (MAGIC) guidelines. Adverse events and SAEs will be assessed from the time of consent through 30 to 35 days after the EOT as per National Cancer Institute CTCAE v4.03. Subjects will be assessed for efficacy (including overall response, NRM, FFS, DOR, relapse rate, relapse-related mortality rates, and OS), safety (including AEs, SAEs, and clinical/laboratory assessments),

#### **Study Population:**

Subjects who have developed Grades II to IV steroid-refractory acute GVHD may be eligible candidates for this study.

#### **Key Inclusion Criteria:**

- · Male or female, 12 years of age or older.
- Have undergone first allogeneic hematopoietic stem cell transplantation (allo-HSCT) from any donor source using bone marrow, peripheral blood stem cells, or cord blood for hematologic malignancies. Recipients of nonmyeloablative and myeloablative conditioning regimens are eligible.

- Clinically suspected Grades II to IV acute GVHD as per MAGIC guidelines, occurring after allogeneic
  hematopoietic stem cell transplant with any conditioning regimen and any anti-GVHD prophylactic
  program. Biopsies should be obtained to pathologically confirm acute GVHD; in cases where a biopsy
  is negative, is unable to be obtained, or is clinically contraindicated, clinical suspicion of acute GVHD
  by the treating physician is sufficient, provided that alternative diagnoses of drug effects or infection are
  adequately ruled out.
- Subjects with steroid-refractory acute GVHD, defined as any of the following:
  - Subjects with progressive GVHD (ie, increase in stage in any organ system or any new organ involvement) after 3 days of primary treatment with methylprednisolone ≥ 2 mg/kg per day (or equivalent).
  - Subjects with GVHD that has not improved (ie, decrease in stage in at least 1 involved organ system) after 7 days of primary treatment with methylprednisolone ≥ 2 mg/kg per day (or equivalent).
  - Subjects who previously began corticosteroid therapy at a lower dose (at least 1 mg/kg per day methylprednisolone) for treatment of skin GVHD or skin GVHD accompanied by upper gastrointestinal (GI) GVHD, but develop new GVHD in another organ system.
  - Subjects who cannot tolerate a corticosteroid taper, that is, begin corticosteroids at 2.0 mg/kg per day, demonstrate response, but progress before a 50% decrease from the initial starting dose of corticosteroids is achieved.
- Evidence of myeloid engraftment (eg, absolute neutrophil count ≥ 0.5 × 10<sup>9</sup>/L for 3 consecutive days if ablative therapy was previously used). Use of growth factor supplementation is allowed.
- Be willing to avoid pregnancy or fathering children based on 1 of the following criteria:
  - Women of nonchildbearing potential (ie, surgically sterile with a hysterectomy and/or bilateral oophorectomy OR ≥ 12 months of amenorrhea).
  - Woman of childbearing potential who has a negative serum pregnancy test at screening and who agrees to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening through safety follow-up. Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the subject and their understanding confirmed.
  - Man who agrees to take appropriate precautions to avoid fathering children (with at least 99% certainty) from screening through safety follow-up. Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the subject and their understanding confirmed.
- Written informed consent and/or assent from the subject, parent, or guardian.
- Willingness to comply with all study visits and procedures.

#### **Key Exclusion Criteria:**

- Has received more than 1 allo-HSCT.
- Has received more than 1 systemic treatment in addition to corticosteroids for acute GVHD.
- Presence of GVHD overlap syndrome as per NIH guidelines.
- Presence of an active uncontrolled infection. An active uncontrolled infection is defined as
  hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs, or
  radiographic findings attributable to infection. Persisting fever without signs or symptoms will not be
  interpreted as an active uncontrolled infection.
- · Known human immunodeficiency virus infection.
- Active hepatitis B virus (HBV) or hepatitis C virus infection that requires treatment or at risk for HBV reactivation. At risk for HBV reactivation is defined as hepatitis B surface antigen positive or antihepatitis B core antibody positive. Previous test results obtained as part of standard of care before allo-HSCT that confirm a subject is immune and not at risk for reactivation (ie, hepatitis B surface antigen negative, surface antibody positive) may be used for purposes of eligibility and tests do not need to be repeated. Subjects with previous positive serology results must have negative polymerase chain

reaction results. Subjects whose immune status is unknown or uncertain must have results confirming immune status before enrollment.

- Serum creatinine > 2.0 mg/dL or creatinine clearance < 40 mL/min measured or calculated by Cockroft-Gault equation.
- Subjects with evidence of relapsed primary disease, or subjects who have been treated for relapse after the allo-HSCT was performed.
- Unresolved toxicity or complications (other than acute GVHD) due to previous allo-HSCT.
- Any corticosteroid therapy for indications other than GVHD at doses of methylprednisolone or equivalent > 1 mg/kg per day within 7 days of enrollment.
- Severe organ dysfunction unrelated to underlying GVHD, including:
  - Cholestatic disorders or unresolved veno-occlusive disease of the liver (defined as persistent bilirubin abnormalities not attributable to GVHD and ongoing organ dysfunction).
  - Clinically significant or uncontrolled cardiac disease, including unstable angina, acute myocardial
    infarction within 6 months from Day 1 of study drug administration, New York Heart Association
    Class III or IV congestive heart failure, circulatory collapse requiring vasopressor or inotropic
    support, or arrhythmia that requires therapy.
  - Clinically significant respiratory disease that requires mechanical ventilation support or 50% oxygen.
- · Currently breast feeding.
- Received Janus kinase (JAK) inhibitor therapy after allo-HSCT for any indication. Treatment with a JAK inhibitor before allo-HSCT is permitted.
- Treatment with any other investigational agent, device, or procedure, within 21 days (or 5 half-lives, whichever is greater) of enrollment. Subjects participating in a GVHD prophylaxis study or conditioning regimen should be discussed with the sponsor's medical monitor before enrollment.
- Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the subject; or interfere with interpretation of study data.
- Known allergies, hypersensitivity, or intolerance to any of the study medications, excipients, or similar compounds.

## Study Drug, Dosage, and Mode of Administration:

Subjects will begin treatment at ruxolitinib 5 mg BID; the dose may be escalated to 10 mg BID after 3 days if hematologic parameters are stable and no treatment-related toxicity is observed. Subjects may have dose reductions during the course of treatment based on safety and laboratory assessments. The dose of ruxolitinib may be re-escalated if toxicity management thresholds are met or if a subject experiences a GVHD flare and has adequate hematologic parameters. The dose of ruxolitinib may not exceed 10 mg BID. Tapering of ruxolitinib is permitted provided the subject has reached the Day 180 visit, achieved a CR or VGPR, and discontinued corticosteroid therapy for at least 8 weeks.

#### Reference Therapy, Dosage, and Mode of Administration:

Subjects will begin treatment at prednisone 2.5 mg/kg per day orally (PO) or methylprednisolone 2.0 mg/kg per day intravenously (IV). Subjects who previously began corticosteroid therapy at a different dose may remain on that dose if considered appropriate by the treating physician. Corticosteroids should be tapered as per institutional guidelines at a rate that is commensurate with resolution of GVHD manifestations.

If GVHD flares during the taper of corticosteroids, then the dose may be re-escalated at the investigator's discretion and will not be considered treatment failure, as long as the dose does not exceed the initial starting dose. If the dose required exceeds this threshold, or if the flare is unresponsive to increased corticosteroids, or if multiple flares are observed, then the subject will be considered to have experienced treatment failure.

### Study Schedule/Key Study Procedures:

| Assessment | Frequency |
|---|---|
| Consent, medical/disease history | Screening |
| GVHD biopsy (as appropriate) | Screening |
| Pregnancy testing (as appropriate) | Screening and as indicated through EOT |
| Electrocardiogram | Screening and as indicated through EOT |
| Physical exam/vitals/ECOG | Screening; weekly to Day 56, then every 28 days through EOT; Day 100; safety follow-up |
| Hematology/chemistry panel | Screening; weekly to Day 56, then every 28 days through EOT; Day 100; safety follow-up |
| Acute GVHD staging | Screening; weekly to Day 56, then every 28 days through EOT; Days 100, 180, and 365; safety follow-up |
| Chimerism assessment | Screening, as indicated up to EOT |
| PTLD assessment | As indicated up to EOT |
| Steroid dose monitoring | Day 1 through EOT |
| Concomitant/prophylactic/supportive care medications | Screening through 30 days after EOT |
| AEs | Screening through 30 days after EOT |

PTLD = post-treatment lymphoproliferative disorder.

### Acute GVHD Staging and Grading, MAGIC Guidelines

| Stage | Skin<br>(Active Erythema Only) | Liver<br>(Bilirubin) | Upper GI | Lower GI<br>(Stool Output/Day) |
|---|---|---|---|---|
| 0 | No active (erythematous)<br>GVHD rash | < 2 mg/dL | No or intermittent<br>nausea, vomiting, or<br>anorexia | Adult: < 500mL/day or<br>< 3 episodes/day.<br>Child: < 10mL/kg per day or<br>< 4 episodes/day. |
| 1 | Maculopapular rash < 25% BSA | 2-3 mg/dL | Persistent nausea,<br>vomiting, or anorexia | Adult: 500-999 mL/day or 3-4 episodes/day. Child: 10-19.9 mL/kg per day or 4-6 episodes/day. |
| 2 | Maculopapular rash 25%-50%<br>BSA | 3.1-6 mg/dL | - | Adult: 1000-1500 mL/day or 5-<br>7 episodes/day.<br>Child: 20-30 mL/kg per day or<br>7-10 episodes/day. |
| 3 | Maculopapular rash > 50% BSA | 6.1-15 mg/dL | - | Adult: > 1500 mL/day or<br>> 7 episodes/day.<br>Child: > 30 mL/kg per day or<br>> 10 episodes/day. |
| 4 | Generalized erythroderma<br>(> 50%) with bullae | > 15 mg/dL | - | Severe abdominal pain with or<br>without ileus or grossly bloody<br>stool (regardless of stool<br>volume). |

BSA = body surface area.

Overall clinical grade (based on most severe target organ involvement):

Grade 0: No Stage 1-4 of any organ.

Grade I: Stage 1-2 skin without liver, upper GI, or lower GI involvement.

Grade II: Stage 3 rash and/or stage 1 liver and/or stage 1 upper GI and/or stage 1 lower GI.

Grade III: Stage 2-3 liver and/or Stage 2-3 lower GI, with Stage 0-3 skin and/or Stage 0-1 upper GI.

Grade IV: Stage 4 skin, liver, or lower GI involvement, with Stage 0-1 upper GI.

**Estimated Duration of Participation:** Subject participation is expected to average 12 months, which includes the following:

- A screening period lasting up to 28 days.
- A treatment period lasting as long as the subject is deriving benefit (estimated 9 months).
- A safety follow-up period lasting 30 to 35 days after treatment ends.
- A survival follow-up period lasting until death, withdrawal of consent, or the end of the study, whichever
  occurs first.

Estimated Number of Subjects: 70

**Estimated Number of Study Sites: 40** 

**Principal Coordinating Investigator: TBD** 

#### Statistical Methods:

Approximately 70 subjects are planned for the final analysis of the primary endpoint. A treatment regimen for steroid-refractory GVHD demonstrating an absolute improvement of 20% versus historic data would be considered clinically meaningful. With the assumed true rate of 60%, a sample size of 70 subjects would provide > 90% probability to have a 95% confidence interval with lower limit of  $\geq$  40%. An interim analysis will be performed for futility once 35 subjects complete the Day 28 visit; if the lower boundary is crossed, the study will be terminated.

## TABLE OF CONTENTS

| SYNOPS | IS | 3 |
|---|---|---|
| LIST OF | ABBREVIATIONS | 15 |
| 1. | INTRODUCTION | 18 |
| 1.1. | Overview of Acute Graft-Versus-Host Disease | 18 |
| 1.1.1. | First-Line Treatment of Acute GVHD | 19 |
| 1.1.2. | Treatment for Steroid-Refractory Acute GVHD | 20 |
| 1.2. | Ruxolitinib Background | 21 |
| 1.2.1. | Pharmacology | 21 |
| 1.2.2. | Clinical Studies | 22 |
| 1.3. | Study Rationale | 23 |
| 1.3.1. | Animal Studies in Acute GVHD Models | 23 |
| 1.3.2. | Clinical Experience With JAK Inhibitors for the Treatment of Acute GVHD | 24 |
| 1.3.3. | Rationale for Chosen Endpoints | 25 |
| 1.4. | Potential Risks and Benefits of the Treatment Regimen | 25 |
| 2. | STUDY OBJECTIVES AND ENDPOINTS | 26 |
| 3. | SUBJECT ELIGIBILITY | 27 |
| 3.1. | Subject Inclusion Criteria | 27 |
| 3.2. | Subject Exclusion Criteria | 28 |
| 4. | INVESTIGATIONAL PLAN | 30 |
| 4.1. | Overall Study Design | 30 |
| 4.2. | Measures Taken to Avoid Bias | 30 |
| 4.3. | Number of Subjects | 30 |
| 4.3.1. | Planned Number of Subjects | 30 |
| 4.3.2. | Replacement of Subjects. | 30 |
| 4.4. | Duration of Treatment and Subject Participation | 30 |
| 4.5. | Overall Study Duration | 31 |
| 4.6. | Study Termination | 31 |
| 5. | TREATMENT | 31 |
| 5.1. | Treatment Assignment | 31 |
| 5.1.1. | Subject Numbering and Treatment Assignment | 31 |
| 512 | Randomization | 32 |

| 5.2. | Study Drugs | 32 |
|---|---|---|
| 5.2.1. | Ruxolitinib | 32 |
| 5.2.1.1. | Description and Administration | 32 |
| 5.2.1.2. | Supply, Packaging, and Labeling | 32 |
| 5.2.1.3. | Storage | 32 |
| 5.2.1.4. | Instruction to Subjects for Handling Ruxolitinib | 33 |
| 5.2.2. | Corticosteroids | 33 |
| 5.2.2.1. | Prednisone | 33 |
| 5.2.2.2. | Methylprednisolone | 33 |
| 5.2.2.3. | Administration of Corticosteroids | 34 |
| 5.2.2.4. | Prophylactic and Supportive Care Medications | 35 |
| 5.3. | Treatment Compliance | 35 |
| 5.4. | Treatment Interruptions and Adjustments | 35 |
| 5.4.1. | Dose Modifications | 35 |
| 5.4.2. | Criteria and Procedures for Dose Interruptions and Adjustments of Ruxolitinib | 35 |
| 5.4.2.1. | Dose Interruptions and Reductions | 35 |
| 5.4.2.2. | Dose Escalation of Ruxolitinib | 38 |
| 5.4.2.3. | Tapering of Ruxolitinib | 38 |
| 5.4.3. | Criteria and Procedures for Dose Interruptions or Adjustments of Corticosteroids | 39 |
| 5.4.4. | Criteria for Permanent Discontinuation of Study Treatment | 39 |
| 5.5. | Withdrawal of Subjects From Study Treatment | 39 |
| 5.5.1. | Withdrawal Criteria | 39 |
| 5.5.2. | Withdrawal Procedures | 40 |
| 5.5.3. | Study Completion | 40 |
| 5.6. | Concomitant Medications | 41 |
| 5.6.1. | Permitted Medications | 41 |
| 5.6.2. | Restricted Medications | 41 |
| 5.6.3. | Prohibited Medications | 41 |
| 6. | STUDY ASSESSMENTS | 41 |
| 6.1. | Screening | 44 |
| 6.2. | Treatment | 45 |

| 6.3. | End of Treatment | 45 |
|----------|---------------------------------------------------------|----|
| 6.4. | Follow-Up | 45 |
| 6.4.1. | Safety Follow-Up | 45 |
| 6.4.2. | GVHD Assessment Follow-Up | 45 |
| 6.4.3. | Survival Follow-Up | 45 |
| 6.5. | Unscheduled Visits | 46 |
| 7. | CONDUCT OF STUDY ASSESSMENTS AND PROCEDURES | 46 |
| 7.1. | Administration of Informed Consent Form | 46 |
| 7.2. | Interactive Response Technology Procedure | 46 |
| 7.3. | Demography and Medical History | 46 |
| 7.3.1. | Demographics and General Medical History | 46 |
| 7.3.2. | Disease Characteristics and Treatment History | 46 |
| 7.4. | Prior and Concomitant Medications | 46 |
| 7.5. | Safety Assessments | 47 |
| 7.5.1. | Adverse Events | 47 |
| 7.5.2. | Physical Examination | 47 |
| 7.5.3. | Vital Signs | 47 |
| 7.5.4. | Eastern Cooperative Oncology Group Performance Status | 47 |
| 7.5.5. | Twelve-Lead Electrocardiograms | 48 |
| 7.5.6. | Laboratory Assessments | 48 |
| 7.5.6.1. | Chemistry | 48 |
| 7.5.6.2. | Hematology | 48 |
| 7.5.6.3. | Pregnancy Testing | 48 |
| 7.5.6.4. | Hepatitis Screening | 49 |
| 7.6. | Graft-Versus-Host Disease Assessments | 49 |
| 7.6.1. | Graft-Versus-Host Disease Staging and Grading | 49 |
| | | 50 |
| 7.6.3. | Donor Chimerism | 50 |
| 7.6.4. | Post-Transplant Lymphoproliferative Disorder Assessment | 51 |
| 7.7. | Pharmacokinetic Assessments | |
| 7.7.1. | Blood Sample Collection | 51 |
| 7.7.2. | Bioanalytical Methodology and Analysis | 51 |
| | | 51 |

| 7.9. | Other Study Procedures | 52 |
|----------|----------------------------------------------|----|
| 7.9.1. | Distribution of Subject Reminder Cards | |
| 8. | SAFETY MONITORING AND REPORTING | |
| 8.1. | Adverse Events | |
| 8.1.1. | Definitions | |
| 8.1.2. | Reporting | |
| 8.2. | Laboratory Test Abnormalities | |
| 8.3. | Serious Adverse Events | |
| 8.3.1. | Definitions | |
| 8.3.2. | Reporting | |
| 8.4. | Emergency Unblinding of Treatment Assignment | |
| 8.5. | Pregnancy | |
| 8.6. | Warnings and Precautions | 57 |
| 8.7. | Data Monitoring Committee | 57 |
| 8.8. | Product Complaints | 57 |
| 9. | STATISTICS | 58 |
| 9.1. | Study Populations | 58 |
| 9.2. | Selection of Sample Size | 58 |
| 9.3. | Level of Significance | 58 |
| 9.4. | Statistical Analyses | 59 |
| 9.4.1. | Primary Analyses | 59 |
| 9.4.2. | Secondary Analyses | 59 |
| | | 60 |
| 9.4.4. | Safety Analyses | 60 |
| 9.4.4.1. | Adverse Events | 60 |
| 9.4.4.2. | Clinical Laboratory Tests | 60 |
| 9.4.4.3. | Vital Signs | 61 |
| 9.4.4.4. | Electrocardiograms | 61 |
| 9.4.5. | Pharmacokinetic Analysis | 61 |
| | | 62 |
| 9.5. | Analyses for the Data Monitoring Committee | 62 |
| 9.6. | Interim Analysis | 62 |

| 10. | ETHICAL CONSIDERATIONS AND ADMINISTRATIVE | |
|---|---|---|
| | PROCEDURES | 63 |
| 10.1. | Investigator Responsibilities | 63 |
| 10.2. | Accountability, Handling, and Disposal of Study Drug | 64 |
| 10.3. | Data Management | 65 |
| 10.4. | Data Privacy and Confidentiality of Study Records | 65 |
| 10.5. | Financial Disclosure | 66 |
| 10.6. | Publication Policy | 66 |
| 11. | REFERENCES | 67 |
| APPENDE | X A. INFORMATION REGARDING EFFECTIVENESS OF<br>CONTRACEPTIVE METHODS | 70 |
| APPENDE | X B. MAGIC GUIDELINES FOR STAGING AND GRADING ACUTE GVHD | 71 |
| APPENDE | X C. CYTOCHROME P450 AND P-GLYCOPROTEIN INHIBITORS AND CYTOCHROME P450 INDUCERS | 73 |

## LIST OF TABLES

| Table 1: | Recommended Corticosteroid Administration Table, Days 1 Through 28 | 34 |
|---|---|---|
| Table 2: | Guidelines for Interruption and Restarting of Ruxolitinib | 36 |
| Table 3: | Dose Reduction Levels for Ruxolitinib | 38 |
| Table 4: | Dose Escalation Levels for Ruxolitinib | 38 |
| Table 5: | Schedule of Assessments | 42 |
| Table 6: | Laboratory Assessments | 43 |
| Table 7: | Clinical Laboratory Analytes | 44 |
| Table 8: | ECOG Performance Status Grades | 47 |
| Table 9: | Pharmacokinetic Sample Collection Time and Windows | 51 |
| Table 10: | Criteria for Clinically Notable Vital Sign Abnormalities | 61 |
| Table 11: | Criteria for Clinically Notable Electrocardiogram Abnormalities | 61 |
| | LIST OF FIGURES | |
| Figure 1: | Summary of Studies Evaluating Agents for Initial Therapy of Acute GVHD <sup>a</sup> | 20 |
| Figure 2: | Summary of Studies Evaluating Agents for Second-Line Therapy of Acute GVHD <sup>a</sup> | 21 |
| Figure 3: | Effect of Ruxolitinib on Survival in Mice After Allo-HSCT | 23 |
| Figure 4: | Ruxolitinib Maintains a Beneficial GVT Effect as Determined by Bioluminescence Imaging in the A20 Leukemia Model | 24 |

## LIST OF ABBREVIATIONS

The following abbreviations and special terms are used in this clinical study Protocol.

| Abbreviation | Definition |
|--------------|---------------------------------------------------------------|
| AE | adverse event |
| aGVHD | acute graft-versus-host disease |
| AIHA | autoimmune hemolytic anemia |
| allo-HSCT | allogeneic hematopoietic stem cell transplantation |
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| ANC | absolute neutrophil count |
| AST | aspartate aminotransferase |
| ATG | antithymocyte globulin |
| BID | twice daily |
| BM | bone marrow |
| BOOP | bronchiolitis obliterans-organizing pneumonia |
| BSA | body surface area |
| CI | confidence interval |
| CIBMTR | Center for International Blood and Marrow Transplant Research |
| CFR | Code of Federal Regulations |
| CMV | cytomegalovirus |
| CR | complete response |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CTFG | Clinical Trial Facilitation Group |
| CYP | cytochrome P450 |
| DNA | deoxyribonucleic acid |
| DOR | duration of response |
| ECOG | Eastern Cooperative Oncology Group |
| ECG | electrocardiogram |
| ECP | extracorporeal photopheresis |
| eCRF | electronic case report form |
| EOT | end of treatment |
| FDA | Food and Drug Administration |
| FFS | failure-free survival |
| GCP | Good Clinical Practice |
| GFP | green fluorescent protein |
| GI | gastrointestinal |

| Abbreviation | Definition |
|---|---|
| GVH | graft versus host |
| GVHD | graft-versus-host disease |
| GVT | graft versus tumor |
| HBV | hepatitis B virus |
| HCV | hepatitis C virus |
| HIPAA | Health Insurance Portability and Accountability Act of 1996 |
| IB | Investigator's Brochure |
| IC <sub>50</sub> | half-maximal inhibitory concentration |
| ICF | informed consent form |
| ICH | International Conference on Harmonisation |
| IEC | independent ethics committee |
| IFN-γ | interferon-γ |
| IFN-γR | interferon-γ receptor |
| IL | interleukin |
| IL-2R | interleukin 2 receptor |
| IN | Investigator Notification |
| IRB | institutional review board |
| ITP | idiopathic thrombocytopenic purpura |
| IUD | intrauterine devices |
| IUS | intrauterine hormone-releasing system |
| IV | intravenously |
| IVRS | interactive voice response system |
| JAK | Janus kinase |
| MAGIC | Mount Sinai Acute GVHD International Consortium |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MHC | major histocompatibility |
| MMF | mycophenolate mofetil |
| MPN | myeloproliferative neoplasm |
| NCI | National Cancer Institute |
| NIH | National Institutes of Health |
| NK | natural killer |
| NR | no response |
| NRM | nonrelapse mortality |
| ORR | overall response rate |
| OS | overall survival |
| PBS | phosphate buffered saline |

| Abbreviation | Definition |
|--------------|----------------------------------------------------|
| PFT | pulmonary function test |
| PK | pharmacokinetic |
| PO | orally |
| PR | partial response |
| PTLD | post-transplant lymphoproliferative disorder |
| QD | once daily |
| RA | rheumatoid arthritis |
| Retro | retrospective |
| RNA | ribonucleic acid |
| SAE | serious adverse event |
| STAT | signal transducers and activators of transcription |
| SUSAR | suspected unexpected serious adverse reaction |
| TEAE | treatment-emergent adverse event |
| TPO | thrombopoietin |
| Treg | regulatory T cell |
| ULN | upper limit of normal |
| VGPR | very good partial response |

#### 1. INTRODUCTION

#### 1.1. Overview of Acute Graft-Versus-Host Disease

Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is an effective immunotherapy for human cancer (Appelbaum 2007). More than 20,000 allo-HSCTs are performed each year worldwide, primarily for the treatment of hematologic malignancies (Pavletic and Fowler 2012). Acute graft-versus-host disease (GVHD) and chronic GVHD remain major contributors to transplantation-related deaths and the most significant barrier to successful allo-HSCT. Graft-versus-host disease occurs when immune cells transplanted from a nonidentical donor (the graft) recognize the transplant recipient (the host) as foreign, thereby initiating an immune reaction that causes disease in the transplant recipient. Despite prophylactic treatments with immunosuppressive agents, approximately 50% of transplantation recipients develop GVHD. Most graft-versus-host (GVH) reactions are undesirable and affect multiple organs; however, GVH reactions against hematopoietic tissue targets are desirable and critical for the cure of hematologic malignancies (ie, the graft-versus-tumor [GVT] effect) and for donor immune-hematopoietic system engraftment. These disparate effects of GVH reactions are difficult to separate, and any strategies directed against GVHD may adversely affect survival by increasing malignancy relapse, graft rejection, and the frequency and severity of infections (Pavletic and Fowler 2012).

There are few therapeutic studies for acute GVHD, and currently no agents are approved by the FDA for either prevention or treatment of acute GVHD (Martin et al 2009). In response to this limitation, an NIH-FDA public workshop was convened in 2009 to facilitate clinical development programs for products to prevent or treat acute GVHD. A major topic of this workshop was defining the optimal endpoint and timing for evaluating new therapeutics for acute GVHD. Although universally accepted as a suitable endpoint for regulatory approval in oncology clinical studies, survival is not always a practical endpoint for developing GVHD therapeutics, owing to the multiple contributing causes of death in the allogeneic transplantation setting (Martin 2008).

Treatment options for GVHD, including modulation of donor-alloreactive effector T-cells, remain a major focus of current therapies for acute GVHD. Other cell populations, including regulatory T cells (Tregs), dendritic cells, natural killer (NK) T cells, and B cells, or other mechanisms, such as modulation of tissue or vascular endothelium damage signals, may also represent targets for GVHD therapy. At diagnosis, the extent of individual organ involvement and overall grade of acute GVHD should be documented, taking into account all organ involvement, as this has prognostic significance. Acute GVHD diagnosis should be confirmed by biopsy of an affected organ if possible; in addition, other non-GVHD complications involving the skin, liver, and gastrointestinal (GI) tract should be ruled out. Although diagnostic biopsies are highly specific if current histopathology criteria are used, the sensitivity of these biopsies is only approximately 60%; therefore, the ultimate acute GVHD diagnosis and decision to treat systemically is based on careful integration of all available clinical information (Weisdorf et al 2003).

The classic target organs for acute GVHD are the skin (severity ranging from maculopapular rash to erythroderma and bullae formation), the GI tract (resulting in nausea, vomiting, abdominal cramps, or diarrhea), and the liver (resulting in hyperbilirubinemia, jaundice, or elevated transaminases). The hematopoietic system can also be targeted, resulting in complete donor lymphohematopoietic chimerism and the GVT response against hematologic malignancies. Endothelium, lungs, and other organs can also be targeted, although skin, gut, and liver involvement are the only organs scored in the current grading system.

The severity of acute GVHD is graded according to the degree of involvement of the skin, liver, and GI tract. Two of the more commonly used grading systems are the Glucksberg system (I-IV) and the International Bone Marrow Transplant Research system (A-D; Glucksberg et al 1974, Rowlings et al 1997). These grading systems have evolved over time, which included refinement of the Glucksberg system by an NIH working group to include persistent nausea with histologic evidence of GVHD as Stage 1 upper GI acute GVHD (Przepiorka et al 1995). The NIH criteria have been further refined by the Mount Sinai Acute GVHD Consortium (MAGIC) to standardize the collection of complex clinical data from multiple organ systems in multicenter studies (Harris et al 2016).

Two subcategories have been recognized within the broader category of acute GVHD: 1) classic acute GVHD (eg, maculopapular erythematous rash, GI symptoms, cholestatic hepatitis), occurring within 100 days after transplantation or donor leukocyte infusion and 2) persistent, recurrent, or late acute GVHD, occurring beyond 100 days after transplantation or donor leukocyte infusion. Both acute GVHD subentities occur without the presence of diagnostic or distinctive chronic GVHD manifestations (Pavletic 2012). The current NIH consensus criteria for assessment of chronic GVHD suggest that clinical manifestations rather than time after transplantation should determine whether the clinical GVHD syndrome is considered acute or chronic (Jagasia et al 2015). Some signs and symptoms are common to both acute GVHD and chronic GVHD (eg, erythema, maculopapular rash, nausea, vomiting or diarrhea, and elevated liver function tests) and thus other characteristics must be used to distinguish between the 2 categories.

#### 1.1.1. First-Line Treatment of Acute GVHD

Corticosteroids are used as conventional first-line systemic therapy, and response rates between 50% and 60% have been previously reported (Saliba et al 2012, MacMillan et al 2010, Levine et al 2010). Treatment with methylprednisone at 2 mg/kg per day (or an oral prednisone equivalent) has been long accepted as standard first-line therapy for acute GVHD in the United States (Martin et al 2012) and Europe (Ruutu et al 2014). In standard-risk cases of upper GI GVHD, reduced doses of systemic corticosteroids (eg, 1 mg/kg per day) and topical steroids have been shown to be equally effective (Mielcarek et al 2009). Neither response rate nor overall survival (OS) advantages were observed in acute GVHD patients treated with corticosteroids at doses higher than 2.5 mg/kg per day (Van Lint et al 1998).

Because only approximately 50% of acute GVHD patients respond to systemic steroids and many of these responses are not durable, attempts have been made to evaluate other agents in addition to prednisone compared with prednisone alone for initial therapy, such as antibodies against interleukin 2 receptor (IL-2R), high-dose steroids, horse antithymocyte globulin, antitumor necrosis factor drugs, mycophenolate mofetil, pentostatin, and sirolimus (Figure 1;

Cahn et al 1995, Lee et al 2004, Cragg et al 2000, Couriel et al 2009, Levine et al 2008, Alousi et al 2009, Pidala et al 2009). In most cases, the second agent yielded modest benefit; however, a study of daclizumab found the additional intervention to be detrimental (Figure 1).

Figure 1: Summary of Studies Evaluating Agents for Initial Therapy of Acute GVHD<sup>a</sup>

| Reference | Agent | Phase | No. of<br>Patients | Response<br>Assessment | CR Proportion | CR or PR<br>Proportion | 6-Month<br>Survival |
|---|---|---|---|---|---|---|---|
| Comparative stu | ıdies | | | | | | |
| [7] | High-dose pred<br>Pred | 3 | 48<br>47 | | | | 0.74<br>0.63 |
| [8] | Low-dose pred<br>Pred | Retro | 347<br>386 | | | | 0.77<br>0.69 |
| [9] | Pred short taper<br>Pred long taper | 3 | 14<br>16 | | | | 0.86<br>0.81 |
| [10] | Basiliximab pred<br>Pred | 3 | 35<br>34 | Day 20<br>Day 20 | 0.54<br>0.44 | 0.63<br>0.71 | 0.78<br>0.66 |
| [12] | Horse ATG pred<br>Pred | 3 | 50<br>46 | Day 42<br>Day 42 | | <b>0.27</b> °<br>0.55 | 0.48<br>0.65 |
| [11] | Daclizumab pred<br>Pred | 3 | 53<br>49 | Day 42<br>Day 42 | 0.43<br>0.49 | 0.51<br>0.53 | 0.53°<br>0.76 |
| [13] <sub>p</sub> | Etanercept pred<br>Pred | 2<br>Retro | 61<br>99 | Day 28<br>Day 28 | <b>0.69<sup>c</sup></b><br>0.33 | | 0.69<br>0.55 |
| [14] <sup>b</sup> | Infliximab pred<br>Pred | 3 | 29<br>28 | Day 28<br>Day 28 | 0.55<br>0.54 | | 0.52<br>0.54 |
| Single-arm studi | es MMFd | Pilot | 17 | | | 0.65 | 0.80 |
| [17]<br>[18] <sup>b</sup> | MMF pred<br>Etanercept pred | Pilot<br>2 | 46 | Day 28 | 0.26 | 0.65 | 0.80 |
| [18] <sub>p</sub> | | 2 | 45 | , | 0.60 | 0.78 | 0.71 |
| [18]b | MMF pred Denileukin pred | 2 | 45<br>47 | Day 28<br>Day 28 | 0.53 | 0.60 | 0.71 |
| [18] <sub>p</sub> | Pentostatin pred | 2 | 42 | Day 28 | 0.38 | 0.62 | 0.56 |
| [19] | Sirolimus | Pilot | 10 | Best | 0.50 | 0.02 | 0.50 |
| Results with pre | dnisone | | | | | | |
| [15] | Pred | 3 | 114 | Day 28 | 0.25 | 0.59 | 0.73 |
| [16] | Pred | Retro | 864 | Day 28 | 0.53 | 0.65 | 0.65 |

aGVHD indicates acute graft-versus-host disease; CR, complete response; PR, partial response; pred, prednisone; Retro, retrospective; ATG, antithymocyte globulin; MMF, mycophenolate mofetil.

Source: Martin et al 2012.

## 1.1.2. Treatment for Steroid-Refractory Acute GVHD

If acute GVHD progresses within 3 days or does not improve after 5 to 7 days of initial treatment, it is considered to be steroid refractory, and second-line therapy is warranted (Pavletic and Fowler 2012). There are no FDA-approved agents for steroid-refractory acute GVHD; numerous combination approaches have been studied, but data do not support the recommendation or exclusion of any particular regimen. Very few prospective studies have evaluated second-line therapy for acute GVHD (Figure 2; Martin et al 2012), and interpretation of these studies is hampered by heterogeneity of subject population, small sample sizes, and lack of standardization in the study design (including timing of the response, different response criteria, and absence of validated endpoints). In addition, treatment of steroid-refractory acute GVHD is associated with significant toxicities, high failure rates, and 6-month survival rate of 49%. Agents that have been investigated over the last 2 decades in these studies include low-dose methotrexate, mycophenolate mofetil, extracorporeal photopheresis, IL-2R targeting (ie, basiliximab, daclizumab, denileukin, and diffitox), alemtuzumab, horse antithymocyte globulin, etanercept, infliximab, and sirolimus (Martin et al 2012).

aNonsteroid treatment results that fall outside the 95% confidence interval for the aggregated overall average of all studies are shown in bold. See Figures 1, 2, and 3.

<sup>&</sup>lt;sup>b</sup>Rationale for planned sample size and corresponding power estimates are reported.

<sup>&</sup>lt;sup>c</sup>Statistically significant difference compared to controls, as reported by the study authors.

Figure 2: Summary of Studies Evaluating Agents for Second-Line Therapy of Acute GVHD<sup>a</sup>

| Agent | Phase | No. of<br>Patients | Response<br>Assessment | CR Proportion | CR or PR<br>Proportion | 6-Month<br>Survival |
|---|---|---|---|---|---|---|
| Methotrexate | Retro | 12 | Day 28 <sup>b</sup> | 0.42 | 0.58 | 0.58 |
| MMF | Retro | 13 | Best | 0.15 | 0.46 | 0.66 |
| MMF | Retro | 10 | Best | 0 | 0.60 | 0.77 |
| MMF | Retro | 48 | Best | 0.31 | 0.79 | 0.47 |
| MMF | Retro | 27 | Best | 0.26 | | 0.52 |
| ECP | Retro | 33 | Best <sup>b</sup> | 0.55 | 0.76 | 0.76 |
| ECP | Retro | 23 | Best <sup>b</sup> | 0.48 | 0.48 | 0.57 |
| Basiliximab | 2 | 23 | Day 7 <sup>b</sup> | 0.17 | 0.83 | 0.55 |
| Daclizumab | 2 | 43 | Day 43 | 0.37 | 0.51 | |
| Daclizumab | 2 | 12 | Day 28 <sup>b</sup> | 0.08 | 0.50 | 0.33 |
| Daclizumab | Retro | 57 | Day 43 | 0.33 | 0.54 | 0.28 |
| Inolimomab | 2 | 14 | Best <sup>b</sup> | 0.14 | 0.43 | 0.36 |
| Denileukin diftitox | 1 | 32 | Best | 0.38 | 0.53 | |
| Denileukin diftitox | 2 | 22 | Best | 0.18 | 0.27 | |
| Alemtuzumab | 2 | 18 | Day 28 <sup>b</sup> | 0.33 | 0.83 | 0.71 |
| Alemtuzumab | 2 | 10 | Best <sup>b</sup> | 0.20 | 0.50 | 0 |
| Alemtuzumab | Retro | 18 | Day 56b | 0.28 | 0.62 | 0.61 |
| Horse ATG | Retro | 22 | Day 28 | | 0.18 | |
| Horse ATG | Retro | 58 | Day 21b | 0.07 | 0.28 | 0.17 |
| Horse ATG | Retro | 79 | Day 28 | 0.20 | 0.54 | 0.44 |
| Horse ATG | 2/3 | 47 | Best <sup>b</sup> | 0.32 | 0.57 | 0.45 |
| Horse ATG | 3 | 27 | Best <sup>b</sup> | 0.33 | 0.56 | 0.55 |
| Etanercept | Retro | 13 | Day 56 | 0.38 | 0.46 | 0.77 |
| Infliximab | Retro | 21 | Day 7 <sup>b</sup> | 0.62 | 0.67 | 0.52 |
| Horse ATG + etanercept | Retro | 16 | Bestb | 0.69 | 0.81 | 0.56 |
| Dacliz + etanercept | 2 | 21 | Best <sup>b</sup> | 0.38 | 0.67 | 0.57 |
| Dacliz + infliximab | Retro | 22 | Day 42 <sup>b</sup> | 0.45 | 0.82 | 0.86 |
| Dacliz/inflix/horse ATG | Retro | 12 | Best <sup>b</sup> | 1.00 | 1.00 | 0.73 |
| Sirolimus | Retro | 34 | Best | 0.44 | 0.76 | 0.48 |

aGVHD = acute graft-versus-host disease; ATG = antithymocyte globulin; CR = complete response; ECP = extracorporeal photopheresis; MMF = mycophenolate mofetil; PR = partial response; Retro = retrospective.

Given these data, the choice of a second-line regimen is made based on the outcome of prior treatments, desired toxicity profile, considerations for drug interactions, logistical practicality, costs, and subject and physician preferences. Second-line treatments, especially those associated with suppression of T cells, are associated with increased infection and viral reactivation (including cytomegalovirus [CMV], Epstein-Barr virus, human herpes virus 6, adenovirus, and polyoma).

## 1.2. Ruxolitinib Background

## 1.2.1. Pharmacology

Ruxolitinib is a novel, potent and selective inhibitor of the Janus kinases (JAKs) with selectivity for JAK1 and JAK2 (Quintás-Cardama et al 2010). Ruxolitinib potently inhibits JAK1 and JAK2 (IC $_{50} < 5$  nM), yet it does not significantly inhibit a broad panel of 28 kinases (< 30% inhibition) when tested at 200 nM (approximately  $100 \times$  the average IC $_{50}$  value for JAK1 and JAK2 enzyme inhibition). In cell-based assays relevant to the pathogenesis of myeloproliferative neoplasms (MPNs), such as JAK/signal transducers and activators of

<sup>&</sup>lt;sup>a</sup> Treatment results that fall outside the 95% confidence interval (CI) for the aggregated overall average of all studies are shown in bold.

b The report did not indicate whether absence of further systemic treatment was a criterion for response. In all other reports, subjects who had further systemic treatment were classified as not having a CR or PR.Source: Martin et al 2012.

transcription (STAT) signaling and the growth of cytokine-dependent tumor cell lines, ruxolitinib demonstrates IC<sub>50</sub> values of 80 to 300 nM. This effect is not due to general cytotoxicity, because ruxolitinib (up to 25 µM) had no significant effect on the growth of a cytokine-independent, Breakpoint cluster region-Abelson-driven cell line. In addition, ruxolitinib inhibited JAK/STAT signaling and growth of a cell line expressing the constitutively active JAK2 mutant (JAK2V617F) that has been implicated in the pathogenesis of the majority of Philadelphia chromosome negative MPNs. Ruxolitinib was also tested in cell-based assays relevant to the increased inflammatory cytokine levels observed in MPNs that contribute to MPN-related systemic symptoms. Ruxolitinib potently inhibited interleukin (IL)-23-stimulated IL-22 production in human T cells ( $IC_{50} = 50 \text{ nM}$ ), as well as IL-6, granulocyte-macrophage colony-stimulating factor and thrombopoietin (TPO)-induced STAT3 phosphorylation in human peripheral blood mononuclear cells with IC<sub>50</sub> values < 100 nM. Ruxolitinib also inhibited granulocyte colony-stimulating factor-stimulated STAT3 phosphorylation in human neutrophils (IC<sub>50</sub> =  $28 \pm 9$  nM), as well as TPO-induced STAT3 phosphorylation in human whole blood  $(IC_{50} = 281 \pm 62 \text{ nM})$ . Finally, ruxolitinib inhibited the production of IL-17 in response to IL-23 in T cells and the production of monocyte chemotactic protein-1 in response to IL-6 in peripheral blood mononuclear cells with IC<sub>50</sub> values of < 120 nM (Fridman et al 2011).

Ruxolitinib inhibited splenomegaly in mice resulting from intravenous (IV) inoculation of cells expressing the clinically relevant JAK2V617F mutation (Quintás-Cardama et al 2010). After 3 weeks of treatment, more than 90% of vehicle-treated mice had succumbed to disease while more than 90% of ruxolitinib-treated mice survived. Treatment with ruxolitinib also reduced inflammatory cytokine levels in these mice. The effects of ruxolitinib were also tested in a mouse disease model of polycythemia vera-like disease, based on transplantation of a 1:1 ratio of JAK2 wild-type green fluorescent protein (GFP)-expressing murine bone marrow cells with JAK2V617F-positive murine bone marrow cells, which have a repopulation advantage. In this model, oral ruxolitinib treatment at doses of 30 or 90 mg/kg twice daily (BID) for 21 consecutive days reduced levels of phosphorylated STAT5 (pSTAT5) in the spleen, as well as the spleen size. Ruxolitinib also effectively reduced the red cell parameters (red blood cell count, hemoglobulin, hematocrit, and reticulocyte count) and neutrophil count. The treatment was well-tolerated as assessed by monitoring body weight, and histological assessments of spleen and bone marrow samples post-therapy revealed a decrease of hypercellularity (erythroid and myeloid lineages) in ruxolitinib-treated groups as compared with vehicle-treated animals. However, no significant decrease in the mutant allele burden surrogate readout (percentage of GFP-negative cells, ie, cells expressing JAK2V617F) was observed, as assessed by flow cytometry. Treatment of mice with ruxolitinib in a cytokine-dependent multiple myeloma xenograft model resulted in a dose-dependent suppression of phosphorylated STAT3 and tumor growth. Efficacy was also observed in additional preclinical tumor models representing both hematologic and solid tumors. Taken together, these data indicate that ruxolitinib will be able to inhibit wild-type and mutant JAKs in the clinical setting and are consistent with its observed efficacy in patients with MPNs.

#### 1.2.2. Clinical Studies

As of 22 FEB 2016, more than 8350 patients have received ruxolitinib in company-sponsored studies. In addition, more than 70 interventional or observational studies sponsored by third

parties are ongoing or completed. Additional details regarding the study designs and primary endpoints of these studies are summarized in the ruxolitinib Investigator's Brochure (IB).

## 1.3. Study Rationale

#### 1.3.1. Animal Studies in Acute GVHD Models

To determine the role of JAK/STAT signaling in GVHD, major histocompatibility (MHC)-mismatched allo-HSCT was performed in mice [B6 (H-2<sup>b</sup>) to Balb/c(H-2<sup>d</sup>)]. In this model, interferon γ receptor (IFN-γR) signaling was shown to play a major role in T-cell trafficking to GVHD target organs via CXCR3. Mice transplanted with IFN-γR -/- T cells had improved survival and less clinical GVHD compared with mice transplanted with wild-type T cells. Furthermore, pharmacologic inhibition of interferon signaling with a JAK/STAT signaling inhibitor, ruxolitinib, for 20 days resulted in the decreased expression of CXCR3, reduced GVHD, and improved survival after allo-HSCT in mice (Figure 3; Choi et al 2012).

Figure 3: Effect of Ruxolitinib on Survival in Mice After Allo-HSCT



BM = bone marrow; INCB = ruxolitinib (INCB018424); PBS = phosphate buffered saline. Source: Choi et al 2012.

This effect was shown to be mediated by altered trafficking of T cells to GVHD target organs. The pharmacologic blockade of JAK/STAT signaling in wild-type T-cells using the JAK/STAT-signaling inhibitor, ruxolitinib, resulted in a similar effect to IFN-γR-/- T cells both *in vitro* (reduction of CXCR3 expression in T cells) and *in vivo* (mitigation of GVHD after allo-HSCT). Ruxolitinib also reduced GVHD and preserved the beneficial GVT effect in 2 different mouse MHC-mismatched allo-HSCT models and 2 different mouse leukemia models (lymphoid leukemia and myeloid leukemia; Figure 4; Choi et al 2014). This result was due to an alteration in T-cell trafficking without affecting T-cell expansion. In addition, prolonged administration of ruxolitinib further improved survival after allo-HSCT. These data suggest that pharmacologic inhibition of JAK/STAT signaling might be a promising therapeutic approach to achieve the beneficial antileukemia effect and overcome human leukocyte antigen barriers in allo-HSCT.

Figure 4: Ruxolitinib Maintains a Beneficial GVT Effect as Determined by Bioluminescence Imaging in the A20 Leukemia Model



BM = bone marrow; INCB = ruxolitinib (INCB018424).

Source: Choi et al 2014.

In a separate study, *in vivo* JAK/STAT signaling inhibition improved survival of mice developing acute GVHD and reduced histopathological GVHD grading, serum levels of proinflammatory cytokines, and expansion of alloreactive luc-transgenic T cells (Choi et al 2012).

It was shown that the JAK1/2 inhibitor ruxolitinib impaired differentiation of CD4<sup>+</sup> T cells into interferon  $\gamma$  (IFN- $\gamma$ ) and IL-17A–producing cells and that both T-cell phenotypes are linked to GVHD. Additionally, ruxolitinib treatment in allo-HSCT recipients increased FoxP3<sup>+</sup> Tregs, which are linked to immunologic tolerance.

## 1.3.2. Clinical Experience With JAK Inhibitors for the Treatment of Acute GVHD

Clinical experience with ruxolitinib in patients with steroid-refractory GVHD was initially reported in 6 patients based on a prospective protocol (Spoerl et al 2014). Results were updated in a retrospective analysis of 95 patients with steroid-refractory acute GVHD (n = 54, all Grade III or IV) or steroid-refractory chronic GVHD (n = 41, all moderate or severe) who were treated with ruxolitinib at a dose of 5 to 10 mg BID (Zeiser et al 2015). Of the 45 patients with acute GVHD (all of whom with Grades 3 or 4 disease), an overall response rate (ORR) of 81.5% was reported, including 25 CRs (46.3%). The median time to response was 1.5 weeks (range 1-11) after initiation of ruxolitinib therapy. In addition, a 6-month survival estimate of 79% (67.3%-90.7%, 95% CI) was reported, with a median follow-up time of 26.5 weeks. Graft-versus-host disease relapses were reported in 6.8% (3/44) of patients. A significant decline in levels of IL-6 and soluble IL-2 receptor were observed in 12 of 25 evaluable patients treated at one center. Cytomegalovirus reactivation was observed in 33.3% (18/54) acute GVHD patients and was controlled using antiviral therapy while ruxolitinib treatment continued. Cytopenias were also observed during treatment with ruxolitinib in 55.5% (30/54) patients; however, cytopenias were reported before treatment with ruxolitinib in 51.7% (28/54). Malignancy relapse was reported in 9.3% (5/54).

A Phase 1 clinical study evaluating INCB039110, a potent, selective inhibitor of JAK1, is currently underway.

Overall, these results suggest that inhibition of JAK/STAT signaling is a promising mechanism in the treatment of acute and chronic GVHD. New treatments for the therapy of acute GVHD after allo-HSCT are urgently needed. Novel treatments with agents targeting the JAK-STAT pathway appear to decrease acute GVHD while preserving GVT in murine models by targeting the IFN- $\gamma$  pathway in activated T cells responsible for acute GVHD. The preclinical data with clinical proof-of-principle findings with ruxolitinib provides a strong rationale and justification of further investigating ruxolitinib with standard corticosteroid doses as a treatment option for patients with acute GVHD.

This study will include subjects who are 12 years and older as data from a Phase 1 study in pediatric subjects showed that safety of ruxolitinib was generally favorable and pharmacokinetic (PK) data were comparable to that in adults (Loh et al 2015). Adolescents between the ages of 12 and 18 years comprise approximately 5% of the adult aGVHD population, and standard treatment does not differ between adolescents and adults.

## 1.3.3. Rationale for Chosen Endpoints

As previously described, very few prospective studies have evaluated second-line therapy for GVHD, and interpretation of these studies is hampered by heterogeneity of patient population and lack of standardization in the study design, including timing of the response, absence of validated evaluation of endpoints, and small numbers of patients. Response rates range between 18% to 79%, and treatment of steroid-refractory acute GVHD is associated with significant toxicities, high failure rates, and 6-month survival rate of 49% (Martin et al 2012).

In order to assess whether response is a significant predictor to long-term clinical benefit, Saliba et al (2012) reported Day 28 response as an independent and strongest predictor statistically of nonrelapse mortality (NRM) at 6 months and at 24 months. Patients with a CR or PR by Day 28 after initiation of systemic therapy had a significantly lower 6-month cumulative incidence of NRM (16%) than patients whose acute GVHD did not respond to therapy by Day 28 (48%, P = 0.005). The impact of Day 28 response on 6-month NRM was independent of acute GVHD severity. Levine et al (2008) reported similar findings showing Day 28 response being predictive of NRM and survival at 6 and 9 months. These findings were further supported by MacMillan et al (2012) in a retrospective study of 864 patients that reported Day 28 and 56 responses were similarly effective in predicting 2-year NRM.

## 1.4. Potential Risks and Benefits of the Treatment Regimen

The primary clinical risks with ruxolitinib treatment are the potential sequelae of decreased hematopoietic proliferation attributable to the inhibition of growth factor pathways associated with JAK inhibition. Dose-dependent, reversible thrombocytopenia, anemia, and neutropenia were the most frequent treatment-emergent adverse events (TEAEs) observed during the Phase 3 clinical studies of ruxolitinib in patients with myelofibrosis. Increased rates of infection and anemia are potential risks of myelosuppression. In healthy volunteers, rheumatoid arthritis patients, and patients with pancreatic cancer or hormone-refractory prostate cancer, the effects on hematopoietic proliferation are less pronounced, presumably because of greater bone marrow reserve. The most frequent nonhematologic adverse events (AEs) were mild, reversible increases in alanine aminotransferase (ALT) and aspartate aminotransferase (AST), bruising,

hypercholesterolemia, dizziness, headache, and urinary tract infections. For a comprehensive assessment of the risks of ruxolitinib, refer to the IB.

## 2. STUDY OBJECTIVES AND ENDPOINTS

| Primary Objective | Primary Endpoint |
|---|---|
| Assess the efficacy of ruxolitinib in combination with corticosteroids in subjects with Grades II to IV steroid-refractory acute GVHD. | ORR at Day 28, defined as the proportion of subjects demonstrating a CR, very good partial response (VGPR), or PR. |
| Secondary Objectives | Secondary Endpoints |
| Assess additional response and longer-term efficacy outcomes in the study population. | Key secondary endpoint: Six-month duration of response (DOR), defined as the time from first response until GVHD progression or death. DOR will be assessed when all subjects complete the Day 180 visit. |
| | ORR, defined as the proportion of subjects demonstrating a CR, VGPR, or PR at Days 14, 56, and 100. |
| | Three-month DOR, defined as the time from first response until GVHD progression or death, when all subjects complete the Day 84 visit. |
| | NRM, defined as the proportion of subjects who died due to causes other than malignancy relapse at Months 6, 9, 12, and 24. |
| | Relapse rate, defined as the proportion of subjects whose underlying malignancy relapses. |
| | Relapse-related mortality rate, defined as the proportion of subjects whose malignancy relapses and has a fatal outcome. |
| | Failure-free survival (FFS), defined as the proportion of subjects who are still alive, have not relapsed, have not required additional therapy for acute GVHD, and have not demonstrated signs or symptoms of chronic GVHD, at Month 6. |
| | OS, defined as the time from study enrollment to death due to any cause. |
| Assess the incidence and severity of AEs and serious adverse events (SAEs). | Summaries of clinical safety data (eg, AEs, infections) will be tabulated and listed. |
| Evaluate the PK of ruxolitinib when administered in combination with corticosteroids. | Maximum observed plasma drug concentration ( $C_{max}$ ), minimum observed plasma drug concentration ( $C_{min}$ ), time of maximum observed plasma drug concentration ( $t_{max}$ ), area under the plasma drug concentration versus time curve (AUC), and apparent clearance of study drug from plasma (CL/F). |



#### 3. SUBJECT ELIGIBILITY

Deviations from eligibility criteria are not allowed, because they can potentially jeopardize the scientific integrity of the study, regulatory acceptability, and/or subject safety. Therefore, adherence to the criteria as specified in the Protocol is essential.

## 3.1. Subject Inclusion Criteria

A subject who meets all of the following criteria may be included in the study:

- 1. Male or female, 12 years of age or older.
- Has undergone first allo-HSCT from any donor source (matched unrelated donor, sibling, haploidentical) using bone marrow, peripheral blood stem cells, or cord blood for hematologic malignancies. Recipients of nonmyeloablative and myeloablative transplants are eligible.
- 3. Clinically suspected Grades II to IV acute GVHD as per MAGIC guidelines, occurring after allo-HSCT with any conditioning regimen and any anti-GVHD prophylactic program. Biopsies should be obtained to pathologically confirm acute GVHD; in cases where a biopsy is negative, is unable to be obtained, or is clinically contraindicated, clinical suspicion of acute GVHD by the treating physician is sufficient, provided that alternative diagnoses of drug effects or infection are adequately ruled out.
- 4. Subjects with steroid-refractory acute GVHD, defined as any of the following:
  - a. Subjects with progressive GVHD (ie, increase in stage in any organ system or any new organ involvement) after 3 days of primary treatment with methylprednisolone ≥ 2 mg/kg per day (or equivalent).

- b. Subjects with GVHD that has not improved (ie, decrease in stage in at least 1 involved organ system) after 7 days of primary treatment with methylprednisolone ≥ 2 mg/kg per day (or equivalent).
- c. Subjects who previously began corticosteroid therapy at a lower dose (at least 1 mg/kg methylprednisolone) for treatment of skin GVHD or skin GVHD accompanied by upper GI GVHD, but develop new GVHD in another organ system.
- d. Subjects who cannot tolerate a corticosteroid taper, that is, begin corticosteroids at 2.0 mg/kg per day, demonstrate response, but progress before a 50% decrease from the initial starting dose of corticosteroids is achieved.
- Evidence of myeloid engraftment (eg, absolute neutrophil count [ANC] ≥ 0.5 × 10<sup>9</sup>/L for 3 consecutive days if ablative therapy was previously used). Use of growth factor supplementation is allowed.
- 6. Be willing to avoid pregnancy or fathering children based on 1 of the following criteria:
  - a. Women of nonchildbearing potential (ie, surgically sterile with a hysterectomy and/or bilateral oophorectomy  $OR \ge 12$  months of amenorrhea).
  - b. Woman of childbearing potential who has a negative serum pregnancy test at screening and who agrees to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening through safety follow-up. Permitted methods that are at least 99% effective in preventing pregnancy (see Appendix A) should be communicated to the subject and their understanding confirmed.
  - c. Man who agrees to take appropriate precautions to avoid fathering children (with at least 99% certainty) from screening through safety follow-up. Permitted methods that are at least 99% effective in preventing pregnancy (see Appendix A) should be communicated to the subject and their understanding confirmed.
- 7. Written informed consent and/or assent from the subject, parent or guardian.
- 8. Willingness to comply with all study visits and procedures.

## 3.2. Subject Exclusion Criteria

- 1. Has received more than 1 allo-HSCT.
- 2. Has received more than 1 systemic treatment in addition to corticosteroids for acute GVHD.
- 3. Presence of GVHD overlap syndrome as per NIH guidelines (Jagasia et al 2015).
- 4. Subjects who have had a splenectomy.
- 5. Presence of an active uncontrolled infection. An active uncontrolled infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs, or radiographic findings attributable to infection. Persisting fever without signs or symptoms will not be interpreted as an active uncontrolled infection.
- 6. Known human immunodeficiency virus infection.

- 7. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection that requires treatment or at risk for HBV reactivation. At risk for HBV reactivation is defined as hepatitis B surface antigen positive or anti-hepatitis B core antibody positive. Previous test results obtained as part of standard of care before allo-HSCT that confirm a subject is immune and not at risk for reactivation (ie, hepatitis B surface antigen negative, surface antibody positive) may be used for purposes of eligibility, and tests do not need to be repeated. Subjects with previous positive serology results must have negative polymerase chain reaction results. Subjects whose immune status is unknown or uncertain must have results confirming immune status before enrollment.
- 8. Serum creatinine > 2.0 mg/dL or creatinine clearance < 40 mL/min as measured or calculated by Cockroft-Gault equation.
- 9. Subjects with evidence of relapsed primary disease, or subjects who have been treated for relapse after the allo-HSCT was performed.
- Unresolved toxicity or complications (other than acute GVHD) due to previous allo-HSCT.
- 11. Any corticosteroid therapy for indications other than GVHD at doses of methylprednisolone or equivalent > 1 mg/kg per day within 7 days of enrollment.
- 12. Severe organ dysfunction unrelated to underlying GVHD, including:
  - a. Cholestatic disorders or unresolved veno-occlusive disease of the liver (defined as persistent bilirubin abnormalities not attributable to GVHD and ongoing organ dysfunction).
  - b. Clinically significant or uncontrolled cardiac disease, including unstable angina, acute myocardial infarction within 6 months from Day 1 of study drug administration, New York Heart Association Class III or IV congestive heart failure, circulatory collapse requiring vasopressor or inotropic support, or arrhythmia that requires therapy.
  - Clinically significant respiratory disease that requires mechanical ventilation support or 50% oxygen.
- 13. Currently breast feeding.
- 14. Received JAK inhibitor therapy after allo-HSCT for any indication. Treatment with a JAK inhibitor before allo-HSCT is permitted.
- 15. Treatment with any other investigational agent, device, or procedure, within 21 days (or 5 half-lives, whichever is greater) of enrollment. Subjects participating in a GVHD prophylaxis study or conditioning regimen should be discussed with the sponsor's medical monitor before enrollment.
- 16. Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the subject; or interfere with interpretation of study data.
- 17. Known allergies, hypersensitivity, or intolerance to any of the study medications, excipients, or similar compounds.

### 4. INVESTIGATIONAL PLAN

## 4.1. Overall Study Design

This is an open-label, single-cohort, multicenter Phase 2 study of ruxolitinib in combination with corticosteroids for the treatment of steroid-refractory Grades II to IV acute GVHD. Eligible subjects will begin treatment at ruxolitinib 5 mg BID; if hematologic parameters are stable and no treatment-related toxicity is observed after the first 3 days of treatment, the dose may be increased to 10 mg BID. Ruxolitinib may be tapered after Day 180 provided the subject has achieved a CR or VGPR and corticosteroids have been discontinued for at least 8 weeks. Subjects who are still receiving calcineurin inhibitors or other agents for GVHD prophylaxis at this time may continue to do so at the treating investigator's discretion. Corticosteroids will be administered at a starting dose of 2.0 mg/kg per day (unless otherwise indicated) on Day 1 and will be tapered as appropriate. Subjects will receive study treatment until treatment failure (progression of GVHD, no response, or requiring additional systemic therapy), unacceptable toxicity, or death. Continued use of anti-infective medications, GVHD prophylaxis medications (including calcineurin inhibitors), transfusion support, and topical steroid therapy is permitted.

Severity of GVHD will be assessed from screening through end of treatment (EOT) using the Mount Sinai Acute GVHD International Consortium (MAGIC) guidelines. Adverse events and SAEs will be assessed from the time of consent through 30 to 35 days after the EOT as per National Cancer Institute (NCI) CTCAE v4.03. Subjects will be assessed for efficacy (including overall response, NRM, FFS, DOR, relapse rate, relapse-related mortality rates, and OS), safety (including AEs, SAEs, and clinical/laboratory assessments),

#### 4.2. Measures Taken to Avoid Bias

Acute GVHD response and AEs will be assessed using standardized objective criteria (MAGIC guidelines [Appendix B] and NCI CTCAE v4.03 [2009], respectively).

## 4.3. Number of Subjects

## 4.3.1. Planned Number of Subjects

This study will enroll approximately 70 subjects with steroid-refractory acute GVHD from approximately 40 study sites.

#### 4.3.2. Replacement of Subjects

Not applicable.

## 4.4. Duration of Treatment and Subject Participation

After signing the informed consent form (ICF), screening assessments may be completed over a period of up to 28 days. Each subject enrolled in the study may continue to receive study treatment for as long as benefit is observed and/or treatment withdrawal criteria are not met. If

the subject discontinues study treatment (ie, ruxolitinib and corticosteroids), then the treatment period will end, and the subject will enter the follow-up period (see Section 6.4). The safety follow-up period will last 30 to 35 days, and the survival follow-up period will last until death, withdrawal of consent, or the end of the study, whichever occurs first. Study participation is expected to average approximately 12 months per individual subject.

## 4.5. Overall Study Duration

The study begins when the first subject signs the informed consent. Subjects who are still receiving study treatment at the time of the primary analysis will be permitted to continue on study treatment until treatment withdrawal criteria are met (Section 5.5). All subjects will be followed for survival until death, withdrawal of consent, or the end of the study, whichever occurs first. The study will end and the final analysis will occur once 75% of subjects have achieved 2-year NRM, died or are lost to follow-up, whichever occurs first.

## 4.6. Study Termination

The investigator retains the right to terminate study participation at any time, according to the terms specified in the study contract. The investigator is to notify the institutional review board (IRB)/independent ethics committee (IEC) in writing of the study's completion or early termination, and send a copy of the notification to the sponsor or sponsor's designee and retain 1 copy for the site study regulatory file.

The sponsor may terminate the study electively or if required by regulatory decision. If the study is terminated prematurely, then the sponsor will notify the investigators, the IRBs and IECs, and the regulatory bodies of the decision and reason for termination of the study.

### 5. TREATMENT

## 5.1. Treatment Assignment

## 5.1.1. Subject Numbering and Treatment Assignment

Each subject will be identified in the study by a subject ID number, which is a combination of the site ID and subject number. Site staff should contact the interactive voice response system (IVRS) to obtain the subject ID number during screening.

Site staff will contact the IVRS to enroll the subject and obtain the initial study drug assignment. The investigator or designee will select the assigned bottles of study drug from their stock that correspond to the number provided by the IVRS, record the bottle numbers in the electronic case report form (eCRF), and dispense the study drug to the subject. All subsequent dispensing of study drug should follow this process. Full details will be provided in the IVRS manual.

All subject numbers will be 6 digits; the first 3 digits will be the site number, and the last 3 digits will be the subject's number. This subject number will be maintained throughout the study and will not be reassigned. Subjects who withdraw consent or discontinue from the study after being assigned a subject number will retain their initial number.

For subjects who signed an ICF but are not allocated and for subjects who are allocated but were not treated, refer to the eCRF Completion Guidelines for instruction on which eCRFs to complete.

#### 5.1.2. Randomization

Not applicable.

## 5.2. Study Drugs

#### 5.2.1. Ruxolitinib

## 5.2.1.1. Description and Administration

Ruxolitinib 5 mg tablets are round and white to off-white in color.

Subjects will begin treatment at ruxolitinib 5 mg BID; if hematologic parameters are stable and no treatment-related toxicity is observed after the first 3 days of treatment, the dose may be increased to 10 mg BID. Stable hematologic parameters are defined as the absence of a  $\geq$  50% decrease in platelet counts and/or ANC relative to Day 1. Ruxolitinib may be taken without regard to food except on days when PK samples are drawn; on those days, subjects should be instructed to fast and refrain from taking ruxolitinib until PK samples are collected. See Section 7.7.1 for additional information.

Subjects may have dose reductions or modifications of ruxolitinib during the course of treatment based on AEs, clinical evaluation, and laboratory assessments. See Section 5.4.1 for dose modifications of ruxolitinib.

Subjects are permitted to remain on ruxolitinib treatment until withdrawal from study treatment is considered necessary as per Section 5.5.

### 5.2.1.2. Supply, Packaging, and Labeling

Ruxolitinib will be supplied as 5 mg tablets packaged in 60-count high-density polyethylene bottles. All tablet excipients comply with the requirements of the applicable compendial monographs.

All Incyte investigational product labels will be in the local language and will comply with the legal requirements of each country and will state "Caution: New Drug--Limited by Federal (or United States) law to investigational use."

### **5.2.1.3.** Storage

Bottles of ruxolitinib tablets should be stored at room temperature, 15°C to 30°C (59°F to 86°F).

## 5.2.1.4. Instruction to Subjects for Handling Ruxolitinib

The subject must be instructed in the handling of study drug as follows:

- To store the study drug at room temperature.
- To only remove from the study drug bottle/kit the number of tablets needed at the time of administration.
- Not to remove doses in advance of the next scheduled administration.
- To make every effort to take doses on schedule.
- To report any missed doses.
- To take study drug within 1 hour after completing a meal (morning and evening meal) with a glass of water.
- Not to take another dose if vomiting occurs after taking study drug.
- To keep study drug in a safe place and out of reach of children.
- To bring all used and unused study drug kits to the site at each visit.

#### 5.2.2. Corticosteroids

Either oral prednisone or IV methylprednisolone may be used to begin corticosteroid treatment at the investigator's discretion.

#### 5.2.2.1. Prednisone

#### **5.2.2.1.1. Description**

Prednisone is a white to off-white, odorless, crystalline powder. Tablets are typically white in color and contain lactose monohydrate, magnesium stearate, microcrystalline cellulose, pregelatinized starch, and sodium starch glycolate. Commonly available dose strengths include 1 mg, 2.5 mg, 5 mg, 10 mg, 20 mg, and 50 mg tablets.

## 5.2.2.1.2. Supply, Packaging, and Labeling

Investigators are responsible for ensuring that subjects receive commercially available supplies of prednisone for the duration of the study treatment period. Incyte may provide prednisone where required by applicable law or regulation.

### 5.2.2.1.3. Storage

Prednisone tablets should be stored in accordance with local prescribing information requirements.

### 5.2.2.2. Methylprednisolone

### **5.2.2.2.1. Description**

Methylprednisolone sterile powder is an anti-inflammatory glucocorticoid, which contains methylprednisolone sodium succinate as the active ingredient. Methylprednisolone sodium succinate, USP, is the sodium succinate ester of methylprednisolone, and it occurs as a white or nearly white, odorless hygroscopic, amorphous solid. It is very soluble in water and in alcohol; it is insoluble in chloroform and is very slightly soluble in acetone.

### 5.2.2.2. Supply, Packaging, and Labeling

Investigators are responsible for ensuring that subjects receive commercially available supplies of methylprednisolone for the duration of the study treatment period. Incyte may provide methylprednisolone where required by applicable law or regulation.

## **5.2.2.2.3.** Storage

Methylprednisolone (unreconstituted product or solution) should be stored in accordance with local prescribing information.

#### 5.2.2.3. Administration of Corticosteroids

Subjects will receive prednisone 2.5 mg/kg per day orally (PO) or methylprednisolone 2.0 mg/kg per day IV. Subjects who previously began corticosteroid therapy at a different dose may remain on that dose if considered appropriate by the treating physician. Corticosteroids should be tapered as per institutional guidelines at a rate that is commensurate with resolution of GVHD manifestations.

A recommended tapering schedule is provided in Table 1.

Table 1: Recommended Corticosteroid Administration Table, Days 1 Through 28

| Study Days | Dose |
|---|---|
| Days 1-5 | Prednisone 2.5 mg/kg QD PO (or methylprednisolone 2.0 mg/kg per day IV) |
| Days 6-10 | Prednisone 2.0 mg/kg QD PO (or methylprednisolone 1.6 mg/kg per day IV) |
| Days 11-15 | Prednisone 1.5 mg/kg QD PO (or methylprednisolone 1.2 mg/kg per day IV) |
| Days 16-20 | Prednisone 1.0 mg/kg QD PO (or methylprednisolone 0.8 mg/kg per day IV) |
| Days 21-25 | Prednisone 0.5 mg/kg QD PO (or methylprednisolone 0.4 mg/kg per day IV) |
| Days 26-28 | Prednisone 0.25 mg/kg QD PO (or methylprednisolone 0.2 mg/kg per day IV) |

QD = once daily.

If GVHD flares during the taper of corticosteroids, then the dose may be re-escalated at the investigator's discretion and will not be considered treatment failure, as long as the dose does not exceed the initial starting dose. If the dose required exceeds this threshold, or if the flare is unresponsive to increased corticosteroids, or if multiple flares are observed, then the subject will be considered to have experienced treatment failure.

Corticosteroids may be taken or administered without regard to food except on days when PK samples are drawn; on those days, subjects should be instructed to fast and refrain from taking corticosteroids until after PK samples are collected. See Section 7.7.1 for additional information.

### 5.2.2.4. Prophylactic and Supportive Care Medications

Patients who undergo allo-HSCT are at risk for a variety of infections based on the degree of immunosuppression induced by the conditioning regimen before transplant. As such, it is considered routine practice to use antibiotics, anti-infectives, and immunizations as prophylactic therapies (Tomblyn et al 2009). In cases where post-transplant anti-infective prophylaxis measures are necessary, ongoing therapy may continue at the investigator's discretion per institutional guidelines.

Systemic and topical GVHD prophylaxis medications (eg, cyclosporine, methotrexate, tacrolimus) may be continued at therapeutic doses as appropriate based on stage and sites of disease.

Additional supportive care measures (eg, use of antimotility agents for diarrhea management) are permitted at the investigator's discretion.

## **5.3.** Treatment Compliance

Compliance with all study-related medications should be emphasized to the subject by the site personnel, and appropriate steps should be taken to optimize compliance during the study. Compliance with ruxolitinib will be calculated by the sponsor based on the drug accountability documented by the site staff and monitored by the sponsor/designee (tablet counts). Subjects will be instructed to bring all study-related medications with them to the study visits in order for site personnel to conduct tablet counts to assess study drug accountability. The drug accountability documentation will be used by the sponsor to calculate treatment compliance.

Although commercial supplies of corticosteroids will be used, dose changes and interruptions will also be documented in the medical record and monitored by the sponsor or its designee. As corticosteroid dose strengths and administration types will vary, compliance with corticosteroids will not be calculated.

## 5.4. Treatment Interruptions and Adjustments

#### 5.4.1. Dose Modifications

Dose interruptions and modifications may occur for individual study subjects based on the presence or absence of toxicity.

### 5.4.2. Criteria and Procedures for Dose Interruptions and Adjustments of Ruxolitinib

#### **5.4.2.1.** Dose Interruptions and Reductions

## 5.4.2.1.1. Toxicity Management

Treatment with ruxolitinib may be delayed up to 14 days to allow for resolution of toxicity (Table 2). Subjects may resume treatment if no medical condition or other circumstance exists that, in the opinion of the investigator, would make the subject unsuitable for further participation in the study. The investigator should contact the sponsor medical monitor to discuss cases where treatment has been delayed for more than 14 days before restarting treatment.

Because subjects may enter the study with compromised bone marrow function, these dose reductions are provided as guidelines; individual decisions regarding dose reduction should be made using clinical judgment and in consultation with the sponsor's medical monitor, taking into account relatedness of the AE to the study drug and the subject's underlying condition. Adverse events that have a clear alternative explanation or transient ( $\leq 72$  hours) abnormal laboratory values without associated clinically significant signs or symptoms may be exempt from dose-reduction rules.

Subjects who are currently receiving ruxolitinib 10 mg BID may be reduced to 5 mg BID; subjects receiving 5 mg BID may be reduced further to 5 mg QD. Subjects who are unable to tolerate ruxolitinib at a dose of 5 mg QD should be withdrawn from study treatment (Table 3).

Table 2: Guidelines for Interruption and Restarting of Ruxolitinib

| Table 2. Guidennes for Interruption and Restarting of Ruxontimo | |
|---|---|
| ADVERSE EVENT | ACTION TAKEN |
| Chemistry | |
| • AST and/or ALT > 3.0 × ULN in subjects with normal ALT/AST at baseline. | <b>Step 1:</b> Interrupt study treatment up to 14 days until the toxicity has resolved to ≤ Grade 1. Exceptions require sponsor approval. |
| | <b>Step 2:</b> Restart study treatment at same dose. If assessed as related to study treatment, restart study treatment at next lower dose and monitor as clinically indicated. |
| | <b>NOTE:</b> In subjects with GVHD-related chemistry elevations at baseline, contact the sponsor medical monitor to discuss clinical management and possible dose reductions. |
| • Total bilirubin elevations that occur in the | • Total bilirubin 3.0–5.0 × ULN: |
| presence of GVHD response that, in the investigator's opinion, cannot be attributed to new liver GVHD or concomitant therapy. | <ul> <li>Repeat assessment within 7 days. If elevation persists: <ul> <li>Reduce ruxolitinib dose by 1 level until bilirubin ≤ 1.5 × ULN.</li> <li>Resume previous dose if resolved in 14 days; if &gt; 14 days, maintain reduced dose.</li> </ul> </li> <li>Total bilirubin &gt;5.0-10.0 × ULN: <ul> <li>Repeat assessment within 7 days. If elevation persists:</li> <li>Hold ruxolitinib until bilirubin ≤ 1.5 × ULN.</li> <li>Monitor LFTs weekly or more frequently as appropriate.</li> <li>Resume previous dose if resolved in 14 days; if &gt; 14 days, resume at reduced dose.</li> </ul> </li> </ul> |
| | <ul> <li>Total bilirubin &gt; 10.0 × ULN: <ul> <li>Repeat assessment within 7 days. If elevation persists:</li> <li>Hold ruxolitinib until bilirubin ≤ 1.5 × ULN.</li> </ul> </li> <li>Resume at reduced dose if resolved in 14 days; if &gt; 14 days, discontinue ruxolitinib and monitor as appropriate.</li> </ul> |
| Total bilirubin elevations that occur in<br>subjects with Stage 1/2 liver GVHD that,<br>in the investigator's opinion, cannot be<br>attributed to worsening liver GVHD or<br>concomitant therapy. | <ul> <li>Total bilirubin &gt; 3.0 × ULN: <ul> <li>Repeat assessment within 7 days. If elevation persists:</li> <li>Reduce ruxolitinib dose by 1 dose level.</li> </ul> </li> <li>If bilirubin ≤ 3.0 × ULN, may resume previous dose.</li> </ul> |
Table 2: Guidelines for Interruption and Restarting of Ruxolitinib (Continued)

| ADVERSE EVENT | ACTION TAKEN |
|---|---|
| Hematology | |
| • ANC < 1.0 × 10 <sup>9</sup> /L, suspected as unrelated to study treatment (eg, GVHD, active CMV viremia). | <ul> <li>Step 1: Reduce dose of ruxolitinib by 1 dose level.</li> <li>Step 2: Monitor ANC count as clinically indicated.</li> <li>Step 3: If ANC count is ≥ 1.0 × 10<sup>9</sup>/L for more than 7 days, then the previous dose of ruxolitinib may be resumed.</li> </ul> |
| <ul> <li>ANC &lt; 1.0 × 10<sup>9</sup>/L, suspected as related to study treatment.</li> <li>ANC &lt; 1.0 × 10<sup>9</sup>/L, with an oral temperature of at least 38.5°C OR with ≥ Grade 3 infection.</li> <li>ANC &lt; 0.5 × 10<sup>9</sup>/L.</li> </ul> | Step 1: Interrupt study treatment for up to 14 days. Step 2: Monitor ANC count as clinically indicated. Step 3: If ANC count is $\geq 1.0 \times 10^9/L$ for more than 7 days, then ruxolitinib may be restarted at 1 dose level below the current dose. Step 4: If ANC count is $\geq 1.0 \times 10^9/L$ for more than 7 days after treatment at a reduced dose, the previous dose level of ruxolitinib may be resumed. |
| • Platelet count is < 10 × 10 <sup>9</sup> /L, or platelet count has decreased by ≥ 50% from baseline, suspected as unrelated to study treatment. | Step 1: Reduce dose of ruxolitinib by 1 dose level. Step 2: Monitor platelet count as clinically indicated. Step 3: If platelet count returns to 20 × 10 <sup>9</sup> /L for more than 7 days, then ruxolitinib may be restarted at 1 dose level below the current dose. |
| <ul> <li>Platelet count is &lt; 10 × 10<sup>9</sup>/L, or platelet count has decreased by ≥ 50% from baseline, suspected as related to study treatment.</li> <li>Platelets &lt; 20 × 10<sup>9</sup>/L, with an oral temperature of at least 38.5°C.</li> </ul> | Step 1: Interrupt study treatment for up to 14 days. Step 2: Monitor platelet count as clinically indicated. Step 3a: If platelet count returns to $20 \times 10^9 / L$ for more than 14 days, then the dose of ruxolitinib may be resumed. Step 3b: If platelet count does not return to $< 10 \times 10^9 / L$ and there is no platelet transfusion-independent recovery to above $< 10 \times 10^9 / L$ , then a bone marrow biopsy should be performed. If megakaryocytic hypoplasia and no platelet transfusion-independent recovery are observed within 72 hours, then study treatment should be discontinued. Step 4: If platelet count remains $\ge 20 \times 10^9 / L$ for more than 7 days after treatment at a reduced dose, then the previous dose level of ruxolitinib may be resumed. |
| Other toxicities | |
| Any Grade 1 or Grade 2 toxicity. | Continue treatment and treat the toxicity; monitor as clinically indicated. |
| Any Grade 3 toxicity, if clinically<br>significant and not manageable by<br>supportive care. | <ul> <li>Step 1: Interrupt study treatment up to 14 days until toxicity resolves to ≤ Grade 1.</li> <li>Step 2: Restart study treatment at same dose; if assessed as related to study treatment, then restart study treatment at next lower dose, and monitor as clinically indicated.</li> </ul> |
| Any recurrent Grade 3 toxicity at 5 mg<br>QD dose. | Discontinue study treatment; follow-up per Protocol. Exceptions require sponsor approval. |
| Any other Grade 4 toxicity. | Discontinue study treatment; follow-up per Protocol. |

ULN = upper limit of normal.

**Table 3:** Dose Reduction Levels for Ruxolitinib

| Current Dose | First Dose Reduction | Second Dose Reduction |
|--------------|----------------------|-----------------------|
| 10 mg BID | 5 mg BID | 5 mg QD |
| 5 mg BID | 5 mg QD | Discontinue |

# 5.4.2.1.2. Coadministration With Strong CYP3A4 Inhibitors or Dual CYP2C9/CYP3A4 Inhibitors

Ruxolitinib is mainly eliminated in humans by oxidative metabolism catalyzed predominantly by cytochrome P450 (CYP) 3A4 and CYP2C9 and is not a substrate for transporters including P-glycoprotein (P-gp). Therefore, concomitant medications that inhibit CYP3A4 and CYP2C9 enzymes might increase exposure to ruxolitinib. See Section 5.6 for additional details.

#### 5.4.2.2. Dose Escalation of Ruxolitinib

Subjects will begin treatment at ruxolitinib 5 mg BID; if hematologic parameters are stable and no treatment-related toxicity is observed after the first 3 days of treatment, the dose may be increased to 10 mg BID. Stable hematologic parameters are defined as the absence of a  $\geq$  50% decrease in platelet counts and/or ANC relative to Day 1.

As described in Table 2, subjects who have had a dose reduction of ruxolitinib in order to manage toxicity may resume treatment at the previous dose if hematologic parameters meet the required threshold(s).

Subjects who have previously had a reduction in the dose of ruxolitinib may have their dose re-escalated if a GVHD flare is experienced, provided that hematologic thresholds are described in Table 2 are met. Dose re-escalation levels of ruxolitinib are described in Table 4.

Dose increases may not exceed 10 mg BID.

Table 4: Dose Escalation Levels for Ruxolitinib

| Current Dose | First Dose Escalation | Second Dose Escalation |
|--------------|-----------------------|------------------------|
| 5 mg QD | 5 mg BID | 10 mg BID |
| 5 mg BID | 10 mg BID | - |

#### 5.4.2.3. Tapering of Ruxolitinib

If a subject has achieved CR or VGPR at Day 180, investigators may begin to taper the dose of ruxolitinib by 1 dose level provided corticosteroids have been discontinued for at least 8 weeks following institutional guidelines. Subjects who are still receiving calcineurin inhibitors or other agents for GVHD prophylaxis at this time may continue to do so at the treating investigator's discretion. In addition, subjects must not be experiencing any Grade 2 or higher hematologic toxicity related to ruxolitinib or symptoms of an active infection. Subsequent reductions to the dose of ruxolitinib may occur after an additional 56 days have elapsed provided the aforementioned requirements are still being met.

Investigators wishing to initiate a taper of ruxolitinib at an earlier timepoint may do so upon consultation with and approval from the sponsor's medical monitor.

If GVHD signs/symptoms worsen during the taper of ruxolitinib, the dose may be escalated by 1 dose level as indicated in Table 4; if the subject requires additional systemic therapy (includes restarting of corticosteroids), then the subject would be considered as having progression of disease and would be withdrawn from study treatment.

If subjects completely taper off ruxolitinib and GVHD signs/symptoms reappear at a later time, ruxolitinib therapy may be restarted at the treating investigator's discretion, and the subject would resume the assessment schedule using the original Day 1 as a reference point.

# 5.4.3. Criteria and Procedures for Dose Interruptions or Adjustments of Corticosteroids

Corticosteroid doses should be tapered as per the recommended tapering schedule in Table 1 or as per institutional guidelines; further dose modifications may be made at the treating investigator's discretion.

### 5.4.4. Criteria for Permanent Discontinuation of Study Treatment

The occurrence of an unacceptable toxicity not caused by the underlying disease will be presumed to be related to study drug treatment and will require that the study drug be permanently discontinued. Unacceptable toxicity is defined as follows:

- Occurrence of an AE that is related to treatment with the study drug that, in the
  judgment of the investigator or the sponsor's medical monitor, compromises the
  subject's ability to continue study-specific procedures or is considered to not be in the
  subject's best interest.
- Persistent AE requiring a delay of therapy for more than 14 days, unless a greater delay has been approved by the sponsor.

# 5.5. Withdrawal of Subjects From Study Treatment

The decision to discontinue study treatment will not constitute study completion (see Section 5.5.3). In the event that the decision is made to discontinue study treatment, the treatment period will be considered complete, and the follow-up period will begin.

#### 5.5.1. Withdrawal Criteria

Subjects **must** be withdrawn from study treatment for the following reasons:

- The subject has experienced an unacceptable toxicity.
- Relapse of the underlying malignancy.
- The subject is unable to tolerate ruxolitinib at a dose of 5 mg QD.
- Additional systemic therapy is required for GVHD progression or lack of response, including corticosteroids equal to or greater than the dose used on Study Day 1.
- Further participation would be injurious to the subject's health or well-being, in the investigator's medical judgment.
- The subject becomes pregnant.

- Consent is withdrawn.
- The study is terminated by the sponsor.
- The study is terminated by the local health authority, IRB, or IEC.

A subject **may** be withdrawn from study treatment as follows:

- If, during the course of the study, a subject is found not to have met eligibility
  criteria, then the medical monitor, in collaboration with the investigator, will
  determine whether the subject should be withdrawn from the study.
- If a subject is noncompliant with study procedures or study drug administration in the investigator's opinion, then the sponsor should be consulted for instruction on handling the subject.

#### 5.5.2. Withdrawal Procedures

In the event that the decision is made to permanently discontinue the study drug, the subject will be withdrawn from the study, and the EOT visit should be conducted. Reasonable efforts should be made to have the subject return for a follow-up visit. These visits are described in Section 6. The last date of the last dose of study drug and the reason for subject withdrawal will be recorded in the eCRF.

### If a subject is withdrawn from study treatment:

- The study monitor or sponsor must be notified.
- The reason(s) for withdrawal must be documented in the subject's medical record and in the eCRF.
- The EOT visit should be performed.
- The date of the EOT visit should be registered in the IVRS.
- Subjects must be followed for safety until the time of the follow-up visit or until study drug-related toxicities resolve, return to baseline, or are deemed irreversible, whichever is longest.

If the subject discontinues study treatment and actively withdraws consent for collection of follow-up data (safety follow-up or disease assessment), then no additional data collection should occur; however, subjects will have the option of withdrawing consent for study treatment but continuing in the follow-up period of the study for safety/efficacy assessments.

#### 5.5.3. Study Completion

A subject will be considered as completing the study if they meet any of the following criteria:

- Subject dies and a date of death is available.
- Subject is known to have died; however, the date of death cannot be obtained. (NOTE: Every effort must be made to obtain the date of death.)
- Subject has discontinued study treatment and has withdrawn consent for collection of follow-up anticancer and survival data.

#### **5.6.** Concomitant Medications

#### 5.6.1. Permitted Medications

Concomitant treatments and/or procedures that are required to manage a subject's medical condition (including prophylactic and/or supportive care medications as described in Section 5.2.2.4) during the study will also be recorded in the eCRF.

#### 5.6.2. Restricted Medications

The following medications have restrictions on use during the treatment period of the study:

- Aspirin in doses exceeding 125 mg per day is not permitted. Low-dose aspirin (≤ 125 mg per day) is permitted unless clinically contraindicated.
- Coadministration with strong CYP 3A inhibitors; consider alternative agents with less CYP3A inhibition (Appendix C). Differences in individual sensitivity and variation CYP enzyme inhibition may result in the need for dose reduction of ruxolitinib and/or corticosteroids as appropriate. The sponsor medical monitor may be consulted for advice when using these agents.
- Coadministration with CYP3A4 inducers (Appendix C).
- If concomitant administration of an anticoagulant/antiplatelet medication is indicated, then caution and enhanced monitoring is required. History of thrombocytopenia should be a factor in the choice of anticoagulant and dose.

#### 5.6.3. Prohibited Medications

The following medications are prohibited during the treatment period of the study:

- Any concurrent anticancer therapy (eg, chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, hormonal therapy, or tumor embolization). Use of biologic agents for treatment of noncancer indications is permitted.
- Any secondary GVHD therapy due to insufficient response/progression on study treatment.
- Concomitant use of a JAK inhibitor.
- Initiating therapy with an investigational medication unless otherwise approved by the medical monitor.

#### 6. STUDY ASSESSMENTS

All study assessments will be performed as indicated in the schedule of assessments (see Table 5), and all laboratory assessments will be performed as indicated in Table 6. Table 7 presents a summary of clinical laboratory analytes to be assessed. The order of assessments is suggested by the order of mention within the schedule. See Section 7 for instructions on each assessment. Further details of study procedures and assessments can be found in the study reference manual.

Table 5: **Schedule of Assessments** 

| | | Screening | | | | | | | | tment | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Phase | | _ | | | | _ | | ase <sup>a</sup> | _ | - h | | | | | | Up Phase |
| Item | Section | -28 to -1 | D1 | D3 | <b>D</b> 7 | D14 | D21 | <b>D28</b> | D35 | D42 | D49 | D56 <sup>b</sup> | D100 | D180 | D365 <sup>c</sup> | <b>EOT</b> | Safety <sup>d</sup> | Survival |
| Informed consent | 7.1 | X | | | | | | | | | | | | | | | | |
| Inclusion/exclusion criteria | 3 | X | | | | | | | | | | | | | | | | |
| Contact IVRS | 7.2 | X | X | | | | | X | | | | X | X | | X | X | | X |
| Demography/disease<br>history | 7.3 | X | | | | | | | | | | | | | | | | |
| Prior/concomitant<br>medications | 7.4 | X | | X | | | | | | | х | X | | | | | | |
| Supportive care medications | 5.2.2.4 | Х | | X | | | | | | х | X | | | | | | | |
| AE assessment | 7.5.1 | X | | | | | | | | X | | | | | | X | X | |
| Physical examination | 7.5.2 | X | X | | X | X | X | X | X | X | X | X | X | | X | X | X | |
| Vital signs | 7.5.3 | X | X | | X | X | X | X | X | X | X | X | X | | X | X | X | |
| ECOG performance status | 7.5.4 | X | X | | X | X | X | X | X | X | X | х | X | | X | х | X | |
| 12-lead ECG | 7.5.5 | X | | | • | | | | As in | licated | | • | | | | X | | |
| Acute GVHD grading and response assessment | 7.6.1 | Х | X | | X | x | X | X | X | X | x | х | X | X | X | х | X | |
| Chimerism assessment | 7.6.3 | X | | | | | | | As in | dicated | | | | | | | | |
| PTLD assessment | 7.6.4 | | | As indicated | | | | | | | | | | | | | | |
| Dispense study drug | 5.1 | | X | | | | | X | | | | X | | | X | | | |
| Study drug compliance | 5.3 | | X | | | | | X | | | | X | | | X | X | | |
| Steroid dose monitoring | 5.3 | | | X | | | | | | | | X | | | | | | |
| Survival follow-up | 6.4 | | | | | | | | | | | | | | | | | X <sup>e</sup> |

 $<sup>\</sup>begin{array}{l} ECG = electrocardiogram; \ PTLD = post-transplant \ lymphoproliferative \ disorder. \\ ^a \ A \pm 2\text{-day window is permitted to facilitate scheduling during the treatment phase.} \end{array}$ 

b After Day 56, visits will occur every 28 days and will include all Day 56 assessments.
c The Day 365 visit will also serve as the regularly scheduled visit occurring every 28 days after Day 56 (ie, Day 364).

d Thirty to 35 days after EOT. For subjects withdrawing due to reasons other than GVHD progression, GVHD status should be assessed every 28 days.

<sup>&</sup>lt;sup>e</sup> Every 8 weeks ± 7 days.

Table 6: **Laboratory Assessments** 

| | | Screening<br>Phase | | Treatment<br>Phase <sup>a</sup> | | | | | ЕОТ | Safety<br>Follow Up | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Item | Section | -28 to -1 | D1 <sup>b</sup> | <b>D3</b> | <b>D</b> 7 | D14 | D21 | D28 | D35 | D42 | D49 | D56 <sup>c</sup> | D100 | D180 | D365 <sup>d</sup> | | Follow-Up |
| Chemistry panel | 7.5.6.1 | X | X | X | X | X | X | X | X | X | X | X | X | | X | X | X |
| Hematology | 7.5.6.2 | X | X | X | X | X | X | X | X | X | X | X | X | | X | X | X |
| Hepatitis screening | 7.5.6.4 | X | | | | | | | | | | | | | | | |
| Serum pregnancy test<br>(childbearing females only) | 7.5.6.3 | X | | | | | | | | | X | | | | | | |
| Urine pregnancy test <sup>e</sup><br>(childbearing females only) | 7.5.6.3 | | | X | | | | | | | | | | | | | |
| PK assessment <sup>f</sup> | 7.7 | | X | | X | X | | | | | | | | | | | |
| Correlative study blood collection | 7.8 | X | X | | X | X | | X | | | | $\mathbf{X}^{g}$ | X | X | X | X | |

a A ± 2-day window is permitted to facilitate scheduling during the treatment phase.
 b Day 1 laboratory assessments do not need to be repeated if screening assessments were performed in preceding 7 days.
 c After Day 56, visits will occur every 28 days and will include all Day 56 assessments.

<sup>&</sup>lt;sup>d</sup> The Day 365 visit will also serve as the regularly scheduled visit occurring every 28 days after Day 56 (ie, Day 364).

<sup>&</sup>lt;sup>e</sup> Urine pregnancy tests are only required if medically indicated and should be confirmed with a serum pregnancy test.

Samples to be collected at predose and at 1 hour ± 15 minutes, at 2 hours ± 30 minutes, and between 4 and 8 hours postdose.

g Day 56 only.

**Table 7: Clinical Laboratory Analytes** 

| Serum Chemistries | Hematology <sup>a</sup> | Other |
|---|---|---|
| Albumin | Hematocrit | Serum pregnancy test |
| ALP | Hemoglobin | Urine pregnancy test <sup>b</sup> |
| ALT | Mean corpuscular volume | |
| AST | Platelet count | |
| Bicarbonate | Red blood cell count | |
| Blood urea nitrogen | Reticulocyte count | |
| Calcium | White blood cell count | |
| Chloride | White blood cell differential (5 parts): | Hepatitis Screening Tests |
| Creatinine | Basophils | _ |
| Glucose | Eosinophils | Hepatitis B surface antigen |
| Lactate dehydrogenase | Lymphocytes | Hepatitis B surface antigen antibody |
| Phosphorus | Monocytes | Hepatitis B core antibody |
| Potassium | Neutrophils | Hepatitis C virus antibody |
| Sodium | - | HCV-RNA |
| Total bilirubin | | HBV-DNA |
| Total protein | | אווס י שוות |

ALP = alkaline phosphatase.

## 6.1. Screening

The screening period is the interval between signing the ICF and the day that the subject is enrolled in the study (Day 1). The screening period may not exceed 28 days. Informed consent must be obtained before performing any study-specific procedures that are not considered standard of care. Assessments that are required to demonstrate eligibility may be performed over the course of 1 or more days during this period.

Procedures conducted as part of the subject's routine clinical management (eg, blood count, imaging study) and obtained before signing the ICF may be used for screening or baseline purposes, provided that the procedure meets the Protocol-defined criteria and has been performed in the timeframe of the study. Results from the screening visit evaluations will be reviewed to confirm subject eligibility before enrollment or the administration of study drug. Tests with results that fail eligibility requirements may be repeated once during the screening period if the investigator believes the results to be in error. For screening assessments that are repeated, the most recent available result before enrollment will be used to determine subject eligibility. Treatment should start as soon as possible, but within 2 days after the date of enrollment. Additionally, a subject who fails screening may repeat the screening process 1 time if the investigator believes that there has been a change in eligibility status (eg, following recovery from an infection).

<sup>&</sup>lt;sup>a</sup> Hematology and chemistry assessments will be performed locally.

<sup>&</sup>lt;sup>b</sup> Urine pregnancy tests are only required if medically indicated.

#### **6.2.** Treatment

The treatment period begins on the day that the subject receives the first dose of study drug through the point at which the principal investigator determines that the subject will be permanently discontinued from the study drug. Dates for subsequent study visits will be determined based on this day and should occur within  $\pm 2$  days of the scheduled date unless delayed for safety reasons. During the Day 1 visit, results from screening visit evaluations should be reviewed to determine whether the subject continues to meet the eligibility requirements as specified in the Protocol.

#### 6.3. End of Treatment

If a decision is made that the subject will permanently discontinue study treatment, then the EOT visit should be conducted. If the EOT visit coincides with a regular study visit, then the EOT evaluations will supersede those of that scheduled visit, and the data should be entered in the EOT visit in the eCRF. The subject should be encouraged to return for the follow-up visit.

# 6.4. Follow-Up

## 6.4.1. Safety Follow-Up

The safety follow-up period is the interval between the EOT visit and the scheduled follow-up visit, which should occur 30 to 35 days after the EOT visit (or after the last dose of study drug if the EOT visit was not performed). Adverse events and SAEs must be reported up until at least 30 after the last dose of study drug, the date of the follow-up visit, or until toxicities resolve, return to baseline, or are deemed irreversible, whichever is longer.

#### 6.4.2. GVHD Assessment Follow-Up

Subjects who discontinue study treatment for reasons other than progression of GVHD will move into the disease status follow-up period and should be assessed every 28 days to monitor disease status. Every effort should be made to collect information regarding disease status until one of the following occurs:

- GVHD progression
- Relapse of malignancy
- Death
- End of study

# 6.4.3. Survival Follow-Up

Once a subject has confirmed GVHD progression or starts a new GVHD therapy, the subject moves into the survival follow-up period and should be contacted by telephone, email, or visit at least every 8 weeks ( $\pm$  7 days) to assess for new GVHD therapy and survival status until death, withdrawal of consent, or the end of the study, whichever occurs first.

## 6.5. Unscheduled Visits

Unscheduled visits may be held at any time at the investigator's discretion, and appropriate clinical and laboratory measurements performed based on AEs or other findings.

#### 7. CONDUCT OF STUDY ASSESSMENTS AND PROCEDURES

#### 7.1. Administration of Informed Consent Form

Valid informed consent must be obtained from the study subject before conducting any study-specific procedures using an ICF approved by the local IRB/IEC that contains all elements required by ICH E6 and describes the nature, scope, and possible consequences of the study in a form understandable to the study subject. Local and institutional guidelines for ICF content and administration must be followed; the original signed ICF must be retained by the investigator, and a copy of the signed ICF must be provided to the study subject. The informed consent process for each subject must be documented in writing within the subject source documentation. Subjects of childbearing potential must agree to take appropriate measures to avoid pregnancy in order to participate in the study (see Appendix A).

# 7.2. Interactive Response Technology Procedure

The IVRS will be contacted to obtain a subject ID number when a subject enters the screening phase. Upon determining that the subject is eligible for study entry, the IVRS will be contacted to obtain study drug assignment. Additionally, the IVRS will be contacted every 28 days to update study drug supply. See Section 5.1.1 for additional information.

# 7.3. Demography and Medical History

# 7.3.1. Demographics and General Medical History

Demographic data and a complete medical and medication history will be collected at screening.

## 7.3.2. Disease Characteristics and Treatment History

A disease-targeted medical and medication history including hematologic malignancy type, current GVHD staging, date of diagnosis, sites of disease, prior anticancer therapy, ablation therapy, prophylaxis therapy, donor type, and other details related to the disease under study will be collected at screening.

#### 7.4. Prior and Concomitant Medications

Prior and concomitant medications will be reviewed to determine subject eligibility. All concomitant medications and measures must be recorded in the eCRF, and any medication received or procedure performed within 30 days before enrollment and up to the end of study will be recorded in the eCRF. The medication record will be maintained after signing the ICF to document concomitant medications, including any changes to the dose or regimen. Concomitant medications include any prescription, over-the-counter, or natural/herbal preparations taken or administered during the study period. Concomitant treatments and/or procedures that are

required to manage a subject's medical condition during the study will also be recorded in the eCRF.

## 7.5. Safety Assessments

#### 7.5.1. Adverse Events

Adverse events will be monitored from the time the subject signs the ICF. Subjects will be instructed to report all AEs during the study and will be assessed for the occurrence of AEs throughout the study. In order to avoid bias in eliciting AEs, subjects will be asked general, nonleading questions such as "How are you feeling?" All AEs (serious and nonserious) must be recorded on the source documents and eCRFs regardless of the assumption of a causal relationship with the study drug. The definition, reporting, and recording requirements for AEs are described in Section 8.

#### 7.5.2. Physical Examination

The targeted physical examination will be a symptom-directed evaluation conducted by the investigator or a medically qualified designee. The targeted physical examination will include assessment(s) of the body systems or organs, as indicated by subject symptoms, AEs, or other findings. Clinically notable abnormalities that are considered clinically significant in the judgment of the investigator are to be reported as AEs.

### 7.5.3. Vital Signs

Vital sign measurements include blood pressure, pulse, respiratory rate, body temperature, and body weight. Blood pressure and pulse will be taken with the subject in the recumbent, semirecumbent, or sitting position. Clinically notable abnormalities that are considered clinically significant in the judgment of the investigator are to be reported as AEs.

#### 7.5.4. Eastern Cooperative Oncology Group Performance Status

Eastern Cooperative Oncology Group performance status (Oken et al 1982; Table 8) will be required at screening and will be assessed at other study visits per Table 5. Performance status must be assessed by a medically qualified individual and recorded in the eCRF.

**Table 8: ECOG Performance Status Grades** 

| Grade | Performance Status |
|---|---|
| 0 | Fully active, able to carry on all predisease performance without restriction. |
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg, light house work, office work. |
| 2 | Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours. |
| 3 | Capable of only limited self-care, confined to bed or chair more than 50% of waking hours. |
| 4 | Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair. |
| 5 | Dead. |

#### 7.5.5. Twelve-Lead Electrocardiograms

A 12-lead ECG will be performed during screening with the subject in a recumbent or semirecumbent position after 5 minutes of rest.

The 12-lead ECG will be interpreted by the investigator at the site and will be used for immediate subject management. The decision to include or exclude a subject or withdraw a subject from the study based on an ECG flagged as "Abnormal, Clinically Significant" is the responsibility of the investigator, in consultation with the sponsor's medical monitor, as appropriate.

Electrocardiograms that are identified as abnormal and clinically meaningful compared with the screening assessment should be reported as AEs. For such AEs, the findings of the abnormal ECGs and the corresponding baseline ECG findings must be reported in the eCRF.

An additional ECG will be performed at the EOT visit; additional ECGs may be performed at the investigator's discretion as clinically indicated.

## 7.5.6. Laboratory Assessments

Blood draws for laboratory assessments will occur at study visits indicated in Table 6. Blood draws will be completed before the subject receives the morning dose of study drug. Specific laboratory assessments are listed in Table 7.

All laboratory assessments will be performed at a local (site) laboratory using institutional best practices. Results and normal reference ranges will be entered into the eCRF.

## **7.5.6.1.** Chemistry

All chemistry assessments will be performed at a local (site) laboratory from blood samples collected using institutional best practices before administration of study drug. Results and normal reference ranges will be entered into the eCRF.

### 7.5.6.2. Hematology

Hematology assessments, including complete blood count with differential, will be performed at a local (site) laboratory using institutional best practices before administration of study drug. Results and normal reference ranges will be entered into the eCRF.

#### 7.5.6.3. Pregnancy Testing

A serum pregnancy test will be required for all women of childbearing potential during screening and at the EOT visit. Urine pregnancy tests will be conducted only if medically indicated. Urine pregnancy tests will be performed locally. If a urine pregnancy test is positive, then the results should be confirmed with a serum pregnancy test.

If the serum pregnancy test is negative after a urine test was positive, then the investigator will assess the potential benefit/risk to the subject and determine whether it is in the subject's best interest to resume study drug and continue participation in the study.

#### 7.5.6.4. Hepatitis Screening

Subjects with active HBV or HCV infection that requires treatment or who are at risk for HBV reactivation are excluded from the study. At risk for HBV reactivation is defined as hepatitis B surface antigen positive or anti-hepatitis B core antibody positive. Prior test results obtained as part of standard of care before allo-HSCT confirming that a subject is immune and not at risk for reactivation (ie, hepatitis B surface antigen negative, surface antibody positive) may be used for purposes of eligibility, and tests do not need to be repeated. Subjects with prior positive serology results must have negative polymerase chain reaction results. Subjects whose immune status is unknown or uncertain must have results confirming immune status before enrollment as per Table 7.

#### 7.6. Graft-Versus-Host Disease Assessments

#### 7.6.1. Graft-Versus-Host Disease Staging and Grading

Acute GVHD grading will be performed by the investigator on a weekly basis for the first 8 weeks after enrollment, then every 28 days thereafter. Graft-versus-host disease staging and grading will also occur on Days 100, 180, and 365 and at the EOT visit. If subjects withdrew due to reasons other than GVHD progression, then GVHD staging and grading will be assessed at the safety follow-up visit. Data regarding the quantification of aGVHD symptoms (extent of skin rash, total bilirubin level, volume of diarrhea) should be reported using MAGIC guidelines (Harris et al 2016); response will be assessed as per the Center for International Blood and Marrow Transplant Research (CIBMTR) modifications to the IBMTR response index as indicated in Appendix B (CIBMTR 2009, Martin et al 2009).

#### Skin:

- Only areas involved with active erythema should be used for determining body surface area staging based on the rule of nines.
- A portion of a body area segment may be used for the quantification.
- Desquamation or fluid-filled bullae should be reported if present as these findings are hallmarks of Stage 4 skin GVHD.

#### Liver:

- Liver GVHD staging is based solely on total (not conjugated/direct) serum bilirubin levels.
- Liver GVHD manifesting as transaminitis without concomitant elevation in serum bilirubin should be diagnosed when the presence of GVHD is confirmed by liver biopsy (where appropriate) and scored as Stage 0.
- If bilirubin levels were elevated before the diagnosis of GVHD in another target organ and do not increase further, then liver GVHD should not be diagnosed in the absence of biopsy confirmation. However, if hyperbilirubinemia develops at the same time or after the onset of GVHD in another target organ, then liver GVHD is presumed to be present in the absence of an identified alternative cause.

# • Upper GI:

- Symptoms of concern for upper GI GVHD include anorexia, nausea, vomiting, and dyspepsia, and assessment depends on close attention to caloric intake and symptom reporting.
- An upper GI endoscopy should be performed whenever possible to confirm upper GI GVHD; however, the diagnosis may be made without biopsy confirmation.
- Graft-versus-host disease is typically not considered as a possible etiology when nausea lasts fewer than 3 days or with fewer than 2 vomiting episodes per day for at least 2 days or anorexia without weight loss.

#### Lower GI:

- Staging of lower GI GVHD relies on accurate measurement of daily stool volumes and documentation of the presence of hematochezia or severe abdominal pain.
- In cases when stool volume cannot be closely measured, volume should be calculated based on an average of 200 mL per episode multiplied by the number of episodes in 24-hour period.
- At the time of GVHD onset, staging should be based on the highest daily volume during the 3 days before diagnosis (excluding volumes attributable to procedures such as bowel preps or endoscopy).
- After the initiation of treatment, lower GVHD staging should be based on the diarrhea volume using (in the order of preference) the following measurements:
   1) average of 3 consecutive days, 2) average of 2 consecutive days, or 3) the volume on day of assessment.
- Severe abdominal pain, ileus, and/or grossly bloody stool should be documented when present, because Stage 4 lower GI GVHD is staged based on the presence of these symptoms and is independent of volume of diarrhea.

#### 7.6.3. **Donor Chimerism**

Donor chimerism after a hematopoietic stem cell transplant involves identifying the genetic profiles of the recipient and of the donor and then evaluating the ratio of donor to recipient cells in the recipient's blood, bone marrow, or other tissue. Chimerism testing using peripheral blood or bone marrow will be performed at the treating investigator's discretion according to local institutional practice as indicated in Table 5. In general, genomic polymorphisms should be assessed via polymerase chain reaction analysis of short tandem repeat loci from isolated lymphocytes or myeloid cells. Fluorescence *in situ* hybridization analysis may also be used in cases with sex-mismatched transplants (Matsuda et al 2004).

### 7.6.4. Post-Transplant Lymphoproliferative Disorder Assessment

Staining for Epstein-Barr virus for PTLD testing will be performed according to local institutional practice at the treating investigator's discretion as indicated in Table 5.

#### 7.7. Pharmacokinetic Assessments

#### 7.7.1. Blood Sample Collection

Pharmacokinetic samples will be obtained on Days 1, 7, and 14. On each of these days, a predose blood sample will be drawn, study treatment will be administered, and serial blood samples will be taken at the intervals shown in Table 9.

The exact date and time of the PK blood draws will be recorded in the eCRF along with the date and time of the last dose of study drug preceding the blood draw (if applicable) and the time of the most recent meal. Instructions for sample preparation and shipping will be provided in the Laboratory Manual. Subjects will receive reminder cards in advance of the study visit providing instruction to hold the dose of study drug on the day of the visit, as well as a place to record the time of the previous dose of study drug and time of the most recent meal or snack consumed.

If PK samples are missing for a subject, PK sample collection should be performed at the next visit. On Days 1, 7, and 14, subjects must refrain from taking study medication before arriving for the visit. Subjects should not have consumed any food within 8 hours before arriving at the clinic. A trough (predose) PK sample (30-minute window) should be drawn at each of the PK visits. Following the trough PK sample, the subject should take the assigned dose of study treatment, and subsequent timed samples will be taken. Food should be withheld until 1 hour after study drug administration.

Table 9: Pharmacokinetic Sample Collection Time and Windows

| Study Day | Timing of Sample Relative to INCB018424 Administration | | | |
|---|---|---|---|---|
| Day 1 | Predose | Predose $ \begin{array}{c c} 1 \text{ h} & 2 \text{ h} \\ \pm 15 \text{ min} & \pm 30 \text{ min} \end{array} $ | | 4-8 h |
| Day 7 | Predose $\begin{array}{c} 1 \text{ h} \\ \pm 15 \text{ m} \end{array}$ | | 2 h<br>± 30 min | 4-8 h |
| Day 14 | Predose | 1 h<br>± 15 min | 2 h<br>± 30 min | 4-8 h |

### 7.7.2. Bioanalytical Methodology and Analysis

Plasma samples will be analyzed for ruxolitinib by a validated liquid chromatography—tandem mass spectrometry assay. These samples will be analyzed by Incyte Corporation (Wilmington, DE) or its designee.

Pharmacokinetic parameters will be calculated from the plasma concentrations of ruxolitinib according to a model-independent approach or population PK approach. Instructions regarding sample collection, handling, and shipping will be provided in the Laboratory Manual.



## 7.9. Other Study Procedures

## 7.9.1. Distribution of Subject Reminder Cards

Subjects will be provided with a reminder card at each visit. The subject reminder card will indicate the date/time of the next visit and will also remind the subject to not take the study drug on Days 1, 7, and 14 until after blood samples for PK and safety have been drawn in the clinic. The reminder cards for the Day 1, 7, and 14 visits will have an area for the subject to record the date and time of the last dose taken (from the previous day) and the time of their last meal before the visit.

## 8. SAFETY MONITORING AND REPORTING

#### **8.1.** Adverse Events

### 8.1.1. Definitions

For the purposes of this Protocol, an adverse event (AE) is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related that occurs after a subject provides informed consent. Abnormal laboratory values or test results occurring after informed consent constitute AEs only if they induce clinical signs or symptoms, are considered clinically meaningful, require therapy (eg, hematologic abnormality that requires transfusion), or require changes in the study drug(s).

#### 8.1.2. Reporting

Adverse events that begin or worsen after informed consent should be recorded on the Adverse Events form of the eCRF. Conditions that were already present at the time of informed consent should be recorded on the Medical History form in the eCRF. Monitoring for the occurrence of new AEs should be continued for at least 30 days after the last dose of study drug. Adverse events (including laboratory abnormalities that constitute AEs) should be described using a diagnosis whenever possible rather than by individual underlying signs and symptoms. When a clear diagnosis cannot be identified, each sign or symptom should be reported as a separate AE.

The term "disease progression" should be recorded as an AE/SAE itself only if there are no other identifiable AEs/SAEs associated with the disease progression at the time of reporting. For events associated with disease progression, the relevant signs and symptoms should be reported using a diagnosis whenever possible rather than individual underlying signs and symptoms. When a clear diagnosis cannot be identified, each sign or symptom should be reported as a separate AE. If the events resulting from disease progression meet the criteria for an SAE (eg, resulted in hospitalization, a life-threatening event, or death), the specific event(s) should be reported as an SAE(s) as described in Section 8.3.2. In both cases (ie, AEs or SAEs related to disease progression), for each event it should be indicated whether the event (diagnosis or signs and symptoms) is related to disease progression.

The severity of AEs will be assessed using CTCAE v4.03 Grades 1 through 4. The CTCAE v4.03 severity of Grade 5 will not be used; AEs resulting in death will be graded accordingly using Grades 1 through 4 and have the outcome noted as fatal. If an event is not classified by CTCAE, the severity of the AE will be graded according to the scale below to estimate the grade of severity:

| Grade 1 | Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. |
|---|---|
| Grade 2 | Moderate; minimally, local, or noninvasive intervention indicated; limiting age-appropriate activities of daily living. |
| Grade 3 | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. |
| Grade 4 | Life-threatening consequences; urgent intervention indicated. |

The occurrence of AEs should be sought by nondirective questioning of the subject during the screening process after signing the ICF and at each visit during the study. Adverse events may also be detected when they are volunteered by the subject during the screening process or between visits, or through physical examination, laboratory test, or other assessments. To the extent possible, each AE should be evaluated to determine:

- The severity grade (CTCAE Grade 1 to 4).
- Whether there is at least a reasonable possibility that the AE is related to the study treatment: suspected (yes) or not suspected (no).
- The start and end dates, unless unresolved at final follow-up.
- The action taken with regard to study drug.
- The event outcome (eg, not recovered/not resolved, recovered/resolved, recovering/resolving, recovered/resolved with sequelae, fatal, unknown).
- The seriousness, as per serious adverse event (SAE) definition provided in Section 8.3.1.

Unlike routine safety assessments, SAEs are monitored continuously and have special reporting requirements (see Section 8.3.2).

All AEs should be treated appropriately. If an AE is treated with a concomitant medication or nondrug therapy, this action should be recorded on Adverse Event form and the treatment should

be specified on the Prior/Concomitant Medications or Procedures and Non-Drug Therapy form in the eCRF.

Once an AE is detected, it should be followed until it has resolved or until it is judged to be permanent; assessment should be made at each visit (or more frequently if necessary) of any changes in severity, the suspected relationship to the study drug, the interventions required to treat the event, and the outcome.

When the severity of an AE changes over time for a reporting period (eg, between visits), each change in severity will be reported as a separate AE until the event resolves. For example, 2 separate AEs will be reported if a subject has Grade 1 diarrhea, meeting the definition of an AE, which lasts for 3 days before worsening to a Grade 3 severity. The Grade 1 event will be reported as an AE with a start date equal to the day the event met the Grade 1 AE definition and a stop date equal to the day that the event increased in severity from Grade 1 to Grade 3. The Grade 3 event will also be reported as an AE, with the start date equal to the day the event changed in intensity from Grade 1 to Grade 3 and a stop date equal to the day that the event either changed severity again or resolved. For analysis purposes, this will be considered 1 AE for this subject, and the highest reported severity will be used.

# 8.2. Laboratory Test Abnormalities

Laboratory abnormalities that constitute an AE in their own right (considered clinically meaningful, induce clinical signs or symptoms, require concomitant therapy, or require changes in study drug) should be recorded on the Adverse Event form in the eCRF. Whenever possible, a diagnosis rather than a symptom should be provided (eg, "anemia" instead of "low hemoglobin"). Laboratory abnormalities that meet the criteria for AEs should be followed until they have returned to normal or an adequate explanation of the abnormality is found. When an abnormal laboratory test result corresponds to a sign or symptom of a previously reported AE, it is not necessary to separately record the laboratory test result as an additional event.

Laboratory abnormalities that do not meet the definition of an AE should not be reported as AEs. A Grade 3 or 4 (severe) AE does not automatically indicate an SAE unless it meets the definition of serious, as defined in Section 8.3.1, and/or per the investigator's discretion. A dose modification for the laboratory abnormality may be required (see Section 5.4.2) and should not contribute to the designation of a laboratory test abnormality as an SAE.

#### 8.3. Serious Adverse Events

## 8.3.1. Definitions

An SAE is defined as an event that meets at least 1 of the following criteria:

- Is fatal or life-threatening.
- Requires inpatient hospitalization or prolongation of existing hospitalization, unless hospitalization is a result of:
  - A routine treatment or monitoring of the studied indication not associated with any deterioration in condition.

- An elective surgery or preplanned treatment for a pre-existing condition that is unrelated to the indication under study and has not worsened since signing the ICF
- A treatment on an emergency outpatient basis for an event not fulfilling any of the definitions of a SAE and not resulting in hospital admission.
- Any social reasons and respite care, in the absence of any deterioration in the subject's general condition.
- Results in persistent or significant disability, incapacity, or a substantial disruption of a person's ability to conduct normal life functions.
- Constitutes a congenital anomaly or birth defect.
- Is considered to be an important medical event or a medically significant event that
  may not result in death, be immediately life-threatening, or require hospitalization but
  may be considered serious when, based upon appropriate medical judgment, the event
  may jeopardize the subject or may require medical or surgical intervention to prevent
  1 of the outcomes listed above.

### 8.3.2. Reporting

Every SAE, regardless of suspected causality (eg, relationship to study drug(s) or study procedure or disease progression), occurring after the subject has signed the ICF through the last study visit (or 30 days) after the last dose of study drug, whichever is later) must be reported to the sponsor (or designee) within **24 hours** of learning of its occurrence, unless otherwise specified by the Protocol. Any SAEs occurring more than 30 days after the last dose of study drug should be reported to the sponsor or its designee only if the investigator suspects a causal relationship to the study drug.

Information about all SAEs is collected and recorded on the Adverse Event form of the eCRF. The investigator must assess and record the causal relationship of each SAE to each specific study drug (ruxolitinib and corticosteroids) during the time it is given.

The investigator must also complete the Incyte Serious Adverse Event Report Form, in English, and send the completed and signed form to the sponsor or designee within 24 hours of becoming aware of the SAE. The investigator must provide a causality assessment, that is, assess whether there is at least a reasonable possibility that the SAE is related to the study treatment: suspected (yes) or not suspected (no). Refer to the Incyte Reference Guide for Completing the Serious Adverse Event Report Form.

The contact information of the sponsor's study-specific representatives is listed in the investigator manual provided to each site. The original copy of the SAE Report Form and the confirmation sheet must be kept at the study site.

Investigational site personnel must report any new information regarding the SAE within 24 hours of becoming aware of the information in the same manner that the initial SAE Report Form was sent. Follow-up information is recorded on an amended or new SAE Report Form, with an indication that it is follow-up to the previously reported SAE and the date of the original report. The follow-up report should include information that was not provided on the previous

SAE Report Form, such as the outcome of the event (eg, resolved or ongoing), treatment provided, action taken with study drug because of the SAE (eg, dose reduced, interrupted, or discontinued), or subject disposition (eg, continued or withdrew from study participation). Each recurrence, complication, or progression of the original event should be reported as follow-up to that event, regardless of when it occurs.

If the SAE is not documented in the IB for the study drug (new occurrence) and is thought to be related to the sponsor's study drug, the sponsor or its designee may urgently require further information from the investigator for reporting to health authorities. The sponsor or its designee may need to issue an Investigator Notification (IN) to inform all investigators involved in any study with the same drug that this SAE has been reported. Suspected Unexpected Serious Adverse Reactions (SUSARs) will be collected and reported to the competent authorities and relevant ethics committees in accordance with Directive 2001/20/EC, or as per national regulatory requirements in participating countries.

# 8.4. Emergency Unblinding of Treatment Assignment

Not applicable.

## 8.5. Pregnancy

Pregnancy, in and of itself, is not regarded as an AE unless there is suspicion that study drug may have interfered with the effectiveness of a contraceptive medication or method. When a pregnancy has been confirmed in a subject during maternal or paternal exposure to study drug, the following procedures should be following in order to ensure subject safety:

- The study drug must be discontinued immediately (female subjects only; see Section 5.4.1 for the maximum permitted duration of study drug interruption).
- The investigator must complete and submit the Incyte Clinical Trial Pregnancy form to the sponsor or its designee within **24 hours** of learning of the pregnancy.

Data on fetal outcome and breastfeeding are collected for regulatory reporting and drug safety evaluation. Follow-up should be conducted for each pregnancy to determine outcome, including spontaneous or voluntary termination, details of the birth, and the presence or absence of any birth defects, congenital abnormalities, or maternal and/or newborn complications, by following until the first well-baby visit. Pregnancy should be recorded on a Clinical Trial Pregnancy form and reported by the investigator to the sponsor or its designee. Pregnancy follow-up information should be recorded on the same form and should include an assessment of the possible causal relationship to the sponsor's study drug to any pregnancy outcome, as well as follow-up to the first well-baby visit or the duration specified in local regulations, whichever is later. Refer to the Incyte Reference Guide for Completing the Clinical Trial Pregnancy Form.

Any SAE occurring during pregnancy must be recorded on the SAE report form and submitted to the sponsor or designee.

## 8.6. Warnings and Precautions

Special warnings or precautions for the study drug, derived from safety information collected by the sponsor or its designee, are presented in the Investigator's Brochure (IB). Additional safety information collected between IB updates will be communicated in the form of Investigator Notifications (INs). Any important new safety information should be discussed with the subject during the study, as necessary. If new significant risks are identified, they will be added to the ICF.

# 8.7. Data Monitoring Committee

There is no formal Data Monitoring Committee review.

The sponsor will continuously monitor safety through frequent contact with the treating investigators, review of the clinical data, and formal study meetings. Routine teleconferences will be held among participating study sites to provide subject-by-subject updates on current study status, interim toxicities reported, and any other pertinent information. Adverse event and laboratory data entered into the clinical database will be reviewed periodically for trends and evolving safety signals.

# 8.8. Product Complaints

The sponsor collects product complaints on study drugs and drug delivery systems used in clinical studies in order to ensure the safety of study participants, monitor quality, and facilitate process and product improvements.

All product complaints associated with material packaged, labeled, and released by the sponsor or its designee will be reported to the sponsor. All product complaints associated with other study material will be reported directly to the respective manufacturer.

The investigator or his/her designee is responsible for reporting a complete description of the product complaint via email or other written communication to the sponsor contact or respective manufacturer as noted in the packaging information. Any AE associated with a product complaint should be reported as described in Section 8.1.2 of this Protocol.

If the investigator is asked to return the product for investigation, he/she will return a copy of the product complaint communication with the product.

#### 9. STATISTICS

# 9.1. Study Populations

Subject enrollment, disposition, demographics, and medical history will be summarized at baseline. Dose exposure will be calculated for each subject. Safety and disease response data will be compared over time to assess change from baseline, during treatment, and follow-up.

The populations to be analyzed include the following:

- Efficacy Evaluable Population: Subjects enrolled into the study.
- Safety Evaluable Population: Subjects enrolled into the study who received at least 1 dose of study drug.
- Pharmacokinetic Evaluable Population: Subjects who receive at least 1 dose of study drug and provide at least 1 plasma sample (1 PK measurement) after study drug administration will be considered as potential PK evaluable subjects. The study pharmacokineticist will review data listings of study drug administration and sample records to identify subjects to be excluded from analyses of PK data.

# 9.2. Selection of Sample Size

Approximately 70 subjects are planned for the final analysis of the primary endpoint of ORR. A treatment regimen for steroid-refractory GVHD demonstrating an absolute improvement of 20% versus historic data would be considered clinically meaningful. With the assumed true rate of 60%, a sample size of 70 subjects would provide > 90% probability to have a 95% CI with lower limit of > 40%.

An interim analysis will be conducted when 35 subjects complete the Day 28 visit in order to assess for futility; if the lower boundary is crossed, the study will be terminated.

A group sequential design method for 1 sample binary outcome data will be used to calculate the lower boundary of futility. The spending function of HSD(-4) will be used. For H0: p = 0.4, Ha: p = 0.6, and a 1-sided binomial test with alpha of 0.025, if  $\leq 15$  subjects respond at the time of the interim analysis, the study will be terminated. This will provide 70.03% probability for the response rate of 40% at the interim analysis.

If  $\geq$  37 subjects respond at the time of final analysis, the study outcome will be considered positive. These assumptions will provide 89.88% power for the response rate of 60% in the final analysis with Type I error of 0.0189.

# 9.3. Level of Significance

No formal statistical tests will be performed. All CIs will be 95%.

# 9.4. Statistical Analyses

## 9.4.1. Primary Analyses

The primary endpoint is ORR at Day 28, defined as the proportion of subjects demonstrating a CR, VGPR, or PR, as per standard criteria (Appendix B). The primary analysis will be conducted once the last subject completes the Day 28 visit or withdraws from the study.

Summary statistics and 95% CI will be provided.

#### 9.4.2. Secondary Analyses

The key secondary endpoint is 6-month DOR, defined as the time from first response until GVHD progression or death. Six-month DOR will be assessed when all subjects complete the the Day 180 visit. The duration of disease control will be estimated by the Kaplan-Meier method.

Additional secondary endpoints will be analyzed as follows:

- ORR, defined as the proportion of subjects demonstrating a CR, VGPR, or PR at Days 14, 56, and 100. Summary statistics and applicable 95% CI will be provided.
- Three-month DOR, defined as the time from first response until GVHD progression or death, when all subjects complete the Day 84 visit.
- NRM, defined as the proportion of subjects who died due to causes other than malignancy relapse at Months 6, 9, 12, and 24. Cumulative incidence rates will be provided. Summary statistics and applicable 95% CI will be provided.
- Relapse rate, defined as the proportion of subjects whose underlying malignancy relapses. The cumulative incidence rate and summary statistics will be provided.
- Relapse-related mortality rate, defined as the proportion of subjects whose
  malignancy relapses and has a fatal outcome. The cumulative incidence rate and
  summary statistics will be provided.
- FFS, defined as the proportion of subjects who are still alive, have not relapsed, have not required additional therapy for acute GVHD, and have not demonstrated signs or symptoms of chronic GVHD, at Month 6. The Kaplan-Meier method will be used. Summary statistics will be provided.
- Overall survival, defined as the time from study enrollment to death due to any cause.
   The Kaplan-Meier method will be used. Summary statistics will be provided.
- Clinical safety data (eg, AEs, infections) will be tabulated and listed.
- The plasma PK of ruxolitinib will be analyzed using a model-independent approach.



#### 9.4.4. Safety Analyses

#### 9.4.4.1. Adverse Events

A TEAE is either any AE reported for the first time or worsening of a pre-existing event after first dose of study drug. Analysis of AEs will be limited to TEAEs, but data listings will include all AEs, regardless of their timing to study drug administration. Adverse events will be tabulated by the MedDRA preferred term and system organ class. Severity of AEs will be based on the NCI CTCAE v4.03.

The subset of AEs considered by the investigator to have a relationship to study drug will be considered to be treatment-related AEs. If the investigator does not specify the relationship of the AE to study drug, then the AE will be considered treatment-related. The incidence of AEs and treatment-related AEs will be tabulated.

#### 9.4.4.2. Clinical Laboratory Tests

Laboratory test values outside the normal range will be assessed for severity based on the normal ranges for the clinical reference laboratory. The incidence of abnormal laboratory values and shift tables relative to baseline will be tabulated.

Laboratory data will be classified into CTC grades for AEs (CTCAE v4.03). The following summaries will be produced for the laboratory data:

 Number and percentage of subjects with worst postbaseline CTC grade (regardless of baseline value) will be summarized. Each subject will be counted only for the worst grade observed postbaseline.

- Shift tables using CTC grades to compare baseline with the worst postbaseline value will be produced with CTC grade.
- For laboratory parameters where CTC grades are not defined, shift tables to the worst
  postbaseline value will be produced using the low/normal/high classifications based
  on laboratory reference ranges.

### **9.4.4.3.** Vital Signs

Descriptive statistics and mean change from baseline will be determined for vital signs (blood pressure, pulse, respiratory rate, and body temperature) at each assessment time. Vital sign results will be reviewed for clinically notable abnormalities (see Table 10), and subjects exhibiting clinically notable vital sign abnormalities will be listed. A value will be considered an "alert" value if it is outside the established range and shows a > 25% change from baseline.

**Table 10:** Criteria for Clinically Notable Vital Sign Abnormalities

| Parameter | High Threshold | Low Threshold |
|--------------------------|----------------|---------------|
| Systolic blood pressure | > 155 mmHg | < 85 mmHg |
| Diastolic blood pressure | > 100 mmHg | < 40 mmHg |
| Pulse | > 100 bpm | < 45 bpm |
| Temperature | > 38°C | < 35.5°C |
| Respiratory rate | > 24/min | < 8/min |

### 9.4.4.4. Electrocardiograms

Descriptive statistics and mean change from baseline will be determined for each ECG parameter at each assessment time. Electrocardiogram results will be reviewed for clinically notable abnormalities according to predefined criteria (Table 11). Subjects exhibiting clinically notable ECG abnormalities will be listed. Adverse events will be reported for clinically notable abnormalities that are considered clinically significant in the judgment of the investigator.

Table 11: Criteria for Clinically Notable Electrocardiogram Abnormalities

| Parameter | High Threshold | Low Threshold |
|-----------|----------------|---------------|
| QTcF | > 460 msec | < 295 msec |
| PR | > 220 msec | < 75 msec |
| QRS | > 120 msec | < 50 msec |
| QT | > 500 msec | < 300 msec |
| RR | > 1330 msec | < 600 msec |

QTcF = Fridericia correction.

#### 9.4.5. Pharmacokinetic Analysis

The PK parameters of C<sub>max</sub>, T<sub>max</sub>, C<sub>min</sub>, AUC<sub>0-t</sub>, and CL/F will be calculated from the blood plasma concentrations of ruxolitinib using standard noncompartmental (model-independent) PK methods. Pharmacokinetic calculations will be performed, if appropriate, using commercial software such as WinNonlin® (Pharsight Corporation, Mountain View, CA). Nominal times will be used in all cases, except when the difference between the actual time and nominal time is greater than 15 minutes for samples collected up to 4 hours after administration and greater than

30 minutes for samples collected more than 4 hours after administration; in these cases, actual time will be used for PK analysis.

If there is a sufficient amount of plasma concentration data from this study, then the data will be analyzed by standard population PK methods using appropriate software (eg, NONMEM).



# 9.5. Analyses for the Data Monitoring Committee

Not applicable.

## 9.6. Interim Analysis

An interim analysis will be conducted when 35 subjects complete Day 28 visit. In this interim analysis, only futility will be assessed, and the study will be terminated if the lower boundary is crossed.

A group sequential design method for 1 sample binary outcome data will be used to calculate the lower boundary of futility. The spending function of HSD(-4) will be used. For H0: p = 0.4, Ha: p = 0.6, and a 1-sided binomial test with alpha of 0.025, if  $\leq 15$  subjects respond at the time of the interim analysis, the study will be terminated. This will provide 70.03% probability for the response rate of 40% at the interim analysis.

If  $\geq$  37 subjects respond at the time of final analysis, the study outcome will be considered positive. These assumptions will provide 89.88% power for the response rate of 60% in the final analysis with Type I error of 0.0189.

# 10. ETHICAL CONSIDERATIONS AND ADMINISTRATIVE PROCEDURES

## 10.1. Investigator Responsibilities

This study will be performed in accordance with ethical principles that originate in the Declaration of Helsinki and conducted in adherence to the study Protocol; GCPs as defined in Title 21 of the US CFR Parts 11, 50, 54, 56, and 312; ICH E6 GCP consolidated guidelines; and local regulatory requirements as applicable to the study locations.

The investigator will be responsible for:

- Permitting study-related monitoring, sponsor audits, IRB/IEC review, and regulatory inspections by providing direct access to source data and other relevant clinical study documents.
  - Monitoring: Qualified representatives of the sponsor or its designee, study
    monitors, will monitor the study according to a predetermined plan. The
    investigator must allow the study monitors to review any study materials and
    subject records at each monitoring visit.
  - Auditing: Qualified representatives of the sponsor or its designee may audit the clinical study site and study data to evaluate compliance with the Protocol, applicable local clinical study regulations, and overall study conduct. The investigator must allow the auditors to review original source records and study documentation for all subjects.
  - Regulatory inspection: Regulatory authorities may conduct an inspection of the study and the site at any time during the development of an investigational product. The investigator and staff are expected to cooperate with the inspectors and allow access to all source documents supporting the eCRFs and other study-related documents. The investigator must immediately notify the sponsor when contacted by any regulatory authority for the purposes of conducting an inspection.
- Obtaining informed consent and ensuring that the study subjects' questions have been answered and the subjects fully understand study procedures:
  - Informed consent must be obtained before any study-related procedures are conducted, unless otherwise specified by the protocol.
  - Informed consent must be obtained using the IRB/IEC-approved version in a language that is native and understandable to the subject. A template will be provided by the sponsor or its designee. The sponsor or its designee must review and acknowledge the site-specific changes to the ICF template. The ICF must include a statement that the sponsor or its designee and regulatory authorities have direct access to subject records.

- Obtaining approval from the IRB/IEC before the start of the study and for any
  changes to the clinical study Protocol, important protocol deviations, routine updates,
  and safety information in accordance with institutional requirements and local law.
  - The investigator is responsible for ensuring that the safety reports provided by the sponsor are reviewed and processed in accordance with regulatory requirements and with the policies and procedures established by the IRB/IEC.
- Adhering to the Protocol as described in this document and agreeing that changes to
  the Protocol procedures, with the exception of medical emergencies, must be
  discussed and approved, first, by the sponsor or its designee and, second, by the
  IRB/IEC. Each investigator is responsible for enrolling subjects who have met the
  specified eligibility criteria.
- Retaining records in accordance with all local, national, and regulatory laws, but for a
  minimum period of at least 2 years after the last marketing application approval in an
  ICH region and until there are no pending or contemplated marketing applications in
  an ICH region, or if not approved, 2 years after the termination of the test article for
  investigation to ensure the availability of study documentation should it become
  necessary for the sponsor or a regulatory authority to review.
  - The investigator must not destroy any records associated with the study without receiving approval from the sponsor. The investigator must notify the sponsor or its designee in the event of accidental loss or destruction of any study records. If the investigator leaves the institution where the study was conducted, the sponsor or its designee must be contacted to arrange alternative record storage options.
  - All eCRF data entered by the site (including audit trail), as well as computer hardware and software (for accessing the data), will be maintained or made available at the site in compliance with applicable record retention regulations. The sponsor will retain the original eCRF data and audit trail.

# 10.2. Accountability, Handling, and Disposal of Study Drug

The investigator is responsible for drug accountability at the study site; however, some of the drug accountability duties may be assigned to an appropriate pharmacist or other designee. Inventory and accountability records must be maintained and readily available for inspection by the study monitor and are open to inspection at any time by any applicable regulatory authorities. The investigator or designee must maintain records that document:

- Delivery of study drug to the study site.
- Inventory of study drug at the site.
- Subject use of the study drug including pill or unit counts from each supply dispensed.
- Return of study drug to the investigator or designee by subjects.

The investigational product must be used only in accordance with the Protocol. The investigator will also maintain records adequately documenting that the subjects were provided the specified

study drug. These records should include dates, quantities, and any available batch or serial numbers or unique code numbers assigned to the investigational product and study subjects.

Completed accountability records will be archived by the site. The investigator or designee will be expected to collect and retain all used, unused, and partially used containers of study drug until verified by the study monitor (unless otherwise agreed to by the sponsor). At the conclusion of the study, the investigator or designee will oversee shipment of any remaining study drug back to the sponsor or its designee for destruction according to institutional standard operating procedures. If local procedures mandate on-site destruction of investigational supply, the site should (where local procedures allow) maintain the investigational supply until the study monitor inspects the accountability records in order to evaluate compliance and accuracy of accountability by the investigative site. At sites where the study drug is destroyed before monitor inspection, the monitors rely on documentation of destruction per the site SOP.

# 10.3. Data Management

Data management will be performed in a validated database via an Electronic Data Capture (EDC) system. All data entry, verification, and validation will be performed in accordance with the current standard operating procedures of the Data Management Department at the sponsor or its designee. The database will be authorized for lock once all defined procedures are completed.

The investigator will be provided with access to an EDC system so that an eCRF can be completed for each subject. Entries made in the eCRF must be verifiable against source documents; if updates to the database are not possible, any discrepancies should be explained and documented. The investigator will be responsible for reviewing all data and eCRF entries and will sign and date the designated forms in each subject's eCRF, verifying that the information is true and correct. The investigator is responsible for the review and approval of all query responses.

Protocol deviations will be identified and recorded in the Protocol Deviation form of the eCRF. The study monitor will reference the Monitoring Plan in order to ensure that each issue identified is appropriately documented, reported, and resolved in a timely manner in accordance with the plan's requirements.

# 10.4. Data Privacy and Confidentiality of Study Records

The investigator and the sponsor, or its designee, must adhere to data privacy laws and regulations. The investigator and the sponsor, or its designee, are responsible for ensuring that sensitive information is handled in accordance with local requirements (eg, HIPAA). Appropriate consent and authorizations for use and disclosure and/or transfer (if applicable) of protected information must be obtained.

Subject names will not be supplied to the sponsor or its designee, if applicable. Only the subject number and subject's initials (subject's initials will only be recorded if allowable by local regulations) will be recorded in the eCRF, where permitted; if the subject's name appears on any other document (eg, laboratory report), it must be obliterated on the copy of the document to be supplied to the sponsor or its designee. Study findings stored on a computer will be stored in accordance with local data protection laws. The subjects will be informed that representatives of the sponsor or its designee, IRB or IEC, or regulatory authorities may inspect their medical

records to verify the information collected, and that all personal information made available for inspection will be handled in strictest confidence and in accordance with local data protection laws.

#### 10.5. Financial Disclosure

Before study initiation, all clinical investigators participating in clinical studies subject to FDA Regulation Title 21 Code of Federal Regulations (CFR) Part 54 – Financial Disclosure by Clinical Investigators (ie, "covered studies") are required to submit a completed Clinical Investigator Financial Disclosure form that sufficiently details any financial interests and arrangements that apply. For the purpose of this regulation, "clinical investigator" is defined as any investigator or subinvestigator who is directly involved in the treatment or evaluation of research subjects, including the spouse and each dependent child of the clinical investigator or subinvestigator. These requirements apply to both US and foreign clinical investigators conducting covered clinical studies.

Any new clinical investigators added to the covered clinical study during its conduct must also submit a completed Investigator Financial Disclosure Form. During a covered clinical study, any changes to the financial information previously reported by a clinical investigator must be reported to the sponsor or its designee. At the conclusion of the covered clinical study, the clinical investigators will be reminded of their obligations. In the event that the clinical investigator is not reminded, they nevertheless will remain obligated to report to the sponsor or its designee any changes to the financial information previously reported, as well as any changes in their financial information for a period of 1 year after completion of the covered clinical study.

# 10.6. Publication Policy

By signing the study Protocol, the investigator and his or her institution agree that the results of the study may be used by the sponsor, Incyte Corporation (Incyte), for the purposes of national and international registration, publication, and information for medical and pharmaceutical professionals. Study results will be published in accordance with applicable local and national regulations. If necessary, the authorities will be notified of the investigator's name, address, qualifications, and extent of involvement. The terms regarding the publication of study results are contained in the agreement signed with the sponsor or its designee. A signed agreement will be retained by the sponsor or its designee.

#### 11. REFERENCES

Alousi AM, Weisdorf DJ, Logan BR, et al. Etanercept, mycophenolate, denileukin, or pentostatin plus corticosteroids for acute graft-versus-host disease: a randomized phase 2 trial from the Blood and Marrow Transplant Clinical Trials Network. Blood 2009;114:511-517.

Appelbaum FR. Hematopoietic-cell transplantation at 50. N Engl J Med 2007;357:1472-1475.

Center for International Blood and Marrow Transplant Research (CIBMTR). Clinical trial endpoints for patients with acute GVHD. 2009.

https://www.cibmtr.org/Meetings/Materials/GVHDworkshop/pages/index.aspx. Accessed February 5, 2015.

Choi J, Cooper, ML, Alahmari B, et al. Pharmacologic blockade of JAK1/JAK2 reduces GvHD and preserves the graft-versus-leukemia effect. PloS One 2014;9:e109799.

Choi J, Ziga ED, Ritchey J, et al. IFNγR signaling mediates alloreactive T-cell trafficking and GVHD. Blood 2012;8:4093-4103.

Cahn JY, Bordigoni P, Tiberghien P, et al. Treatment of acute graft-versus-host disease with methylprednisolone and cyclosporine with or without an anti-interleukin-2 receptor monoclonal antibody: a multicenter phase III study. Transplantation 1995;60:939-942.

Clinical Trial Facilitation Group (CTFG). Recommendations related to contraception and pregnancy testing in clinical trials. 2014. http://www.hma.eu/ctfg.html. Accessed June 8, 2015.

Couriel DR, Saliba R, de Lima M, et al. A phase III study of infliximab and corticosteroids for the initial treatment of acute graft-versus-host disease. Biol Blood Marrow Transplant 2009:15:1555-1562.

Cragg L, Blazar BR, Defor T, et al. A randomized trial comparing prednisone with antithymocyte globulin/prednisone as an initial systemic therapy for moderately severe acute graft-versus-host disease. Biol Blood Marrow Transplant 2000;6:441-447.

Fridman JS, Scherle PA, Collins R, et al. Preclinical evaluation of local JAK1 and JAK2 inhibition in cutaneous inflammation. J Invest Dermatol 2011;131:1838-1844.

Glucksberg H, Storb R, Fefer A, et al. Clinical manifestations of graft-versus-host disease in human recipients of marrow from HL-A-matched sibling donors. Transplantation 1974:18:295-304.

Harris AC, Young R, Devine S, et al. International, Multicenter Standardization of Acute Graft-versus-Host Disease Clinical Data Collection: A Report from the Mount Sinai Acute GVHD International Consortium. Biol Blood Marrow Transplant 2016;22:4-10.

INCB018424 Investigator's Brochure (IB). Wilmington, DE: Incyte Corporation.

Jagasia MH, Greinix HT, Arora M, et al. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: I. The 2014 Diagnosis and Staging Working Group report. Biol Blood Marrow Transplant 2015;21:389-401.

Lee SJ, Zahrieh D, Agura E, et al. Effect of up-front daclizumab when combined with steroids for the treatment of acute graft-versus-host disease: results of a randomized trial. Blood 2004;104:1559-1564.

Levine JE, Logan B, Wu J, et al. Graft-versus-host disease treatment: predictors of survival. Biol Blood Marrow Transplant 2010;16:1693-1699.

Levine JE, Paczesny S, Mineishi S, et al. Etanercept plus methylprednisolone as initial therapy for acute graft-versus-host disease. Blood 2008;111:2470-2475.

Loh ML, Tasian SK, Rabin KR, et al. A phase 1 dosing study of ruxolitinib in children with relapsed or refractory solid tumors, leukemias, or myeloproliferative neoplasms: A Children's Oncology Group phase 1 consortium study (ADVL1011). Pediatr Blood Cancer 2015;62:1717-1724.

MacMillan ML, DeFor TE, Weisdorf DJ. The best endpoint for acute GVHD treatment trials. Blood 2010;115:5412-5417.

MacMillan ML, DeFor TE, Weisdorf DJ. What predicts high risk acute graft-versus-host disease (GVHD) at onset?: identification of those at highest risk by a novel acute GVHD risk score. Br J Haematol 2012;157:732-741.

Maecker HT, McCoy JP, Nussenblatt R. Standardizing immunophenotyping for the Human Immunology Project. Nat Rev Immunol 2012;12:191-200.

Magenau JM, Qin X, Tawara I, et al. Frequency of CD4(+)CD25(hi)FOXP3(+) regulatory T cells has diagnostic and prognostic value as a biomarker for acute graft-versus-host-disease. Biol Blood Marrow Transplant, 2010;16:907-914.

Martin PJ. Study design and endpoints in graft-versus-host disease. Best Pract Res Clin Haematol 2008;21:357-372.

Martin PJ, Bachier CR, Klingemann HG, et al. Endpoints for clinical trials testing treatment of acute graft-versus-host disease: a joint statement. Biol Blood Marrow Transplant 2009;15:777-784.

Martin PJ, Rizzo JD, Wingard JR, et al. First- and second-line systemic treatment of acute graft-versus-host disease: recommendations of the American Society of Blood and Marrow Transplantation. Biol Blood Marrow Transplant 2012;18:1150-1163.

Matsuda K, Yamauchi K, Tozuka M, et al. Monitoring of hematopoietic chimerism by short tandem repeats, and the effect of CD selection on its sensitivity. Clin Chem 2004;50:2411-2414.

Mielcarek M, Storer BE, Boeckh M, et al. Initial therapy of acute graft-versus-host disease with low-dose prednisone does not compromise patient outcomes. Blood 2009;113:2888-2894.

Miyara M, Yoshioka Y, Kitoh A, et al. Functional delineation and differentiation dynamics of human CD4+ T cells expressing the FoxP3 transcription factor. Immunity 2009;30:899-911.

National Cancer Institute (NCI). Common Terminology Criteria for Adverse Events (CTCAE) v4.03. 2009. http://ctep.cancer.gov/reporting/ctc.html. Accessed June 9, 2016.

Oken MM, Creech RH, Tormey DC, et al. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol 1982;5:649-655.

Pavletic SZ. Response as an end point in treatment trials for acute GVHD. Bone Marrow Transplant 2012;47:161-163.

Pavletic SZ, Fowler DH. Are we making progress in GVHD prophylaxis and treatment? Hematology Am Soc Hematol Educ Program 2012;251-264.

Pidala J, Kim J, Anasetti C. Sirolimus as primary treatment of acute graft-versus-host disease following allogeneic hematopoietic cell transplantation. Biol Blood Marrow Transplant 2009;15:881-885.

Przepiorka D, Weisdorf D, Martin P, et al. 1994 Consensus Conference on Acute GVHD Grading. Bone Marrow Transplant 1995;15:825-828.

Quintás-Cardama A, Vaddi K, Liu P, et al. Preclinical characterization of the selective JAK1/2 inhibitor INCB018424: therapeutic implications for the treatment of myeloproliferative neoplasms. Blood 2010;115:3109-3117.

Rowlings PA, Przepiorka D, Klein JP, et al. IBMTR Severity Index for grading acute graft-versus-host disease: retrospective comparison with Glucksberg grade. Br J Haematol 1997;97:855-864.

Ruutu T, Gratwohl A, de Witte T, et al. Prophylaxis and treatment of GVHD: EBMT–ELN working group recommendations for a standardized practice. Bone Marrow Transplant 2014;49:168-173.

Sakaguchi S, Miyara M, Constantino CM, Hafler DA. FOXP3+ regulatory T cells in the human immune system. Nat Rev Immunol 2010;10:490-500.

Saliba RM, Couriel DR, Giralt S, et al. Prognostic value of response after upfront therapy for acute GVHD. Bone Marrow Transplant 2012;47:125-131.

Spoerl S, Maas-Bauer K, Verbeek M, et al. Response to JAK 1/2 inhibition in patients with corticosteroid-refractory acute graft-versus-host disease. Poster presented at: 56th ASH Annual Meeting and Exposition; December 6-9, 2014; San Francisco, CA.

Tomblyn M, Chiller T, Einsele H, et al. Guidelines for preventing infectious complications among hematopoietic cell transplantation recipients: a global perspective. Biol Blood Marrow Transplant 2009;15:1143-1238.

Van Lint MT, Uderzo C, Locasciulli A, et al. Early treatment of acute graft-versus-host disease with high- or low-dose 6-methylprednisolone: a multicenter randomized trial from the Italian Group for Bone Marrow Transplantation. Blood 1998; 92:2288-2293.

Weisdorf DJ, Hurd D, Carter S, et al. Prospective grading of graft-versus-host disease after unrelated donor marrow transplantation: a grading algorithm versus blinded expert panel review. Biol Blood Marrow Transplant 2003;9:512-518.

Zeiser R, Burchert A, Lengerke C, et al. Ruxolitinib in corticosteroid-refractory graft-versus-host disease after allogeneic stem cell transplantation: a multicenter survey. Leukemia 2015;29:2062-2068.

# APPENDIX A. INFORMATION REGARDING EFFECTIVENESS OF CONTRACEPTIVE METHODS

## For Subjects Participating in the Study:

The following methods that can achieve a failure rate of less than 1% per year when used consistently and correctly are considered as highly effective birth control methods.

#### Such methods include:

- Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation<sup>1</sup>
  - oral
  - intravaginal
  - transdermal
- Progestogen-only hormonal contraception associated with inhibition of ovulation<sup>1</sup>
  - oral
  - injectable
  - implantable<sup>2</sup>
- Intrauterine device (IUD)<sup>2</sup>
- Intrauterine hormone-releasing system (IUS)<sup>2</sup>
- Bilateral tubal occlusion<sup>2</sup>
- Vasectomised partner<sup>2,3</sup>
- Sexual abstinence<sup>4</sup>

Source: CTFG 2014.

<sup>&</sup>lt;sup>1</sup> Hormonal contraception may be susceptible to interaction with the IMP, which may reduce the efficacy of the contraception method.

<sup>&</sup>lt;sup>2</sup> Contraception methods that in the context of this guidance are considered to have low user dependency.

<sup>&</sup>lt;sup>3</sup> Vasectomised partner is a highly effective birth control method provided that partner is the sole sexual partner of the WOCBP trial participant and that the vasectomised partner has received medical assessment of the surgical success

<sup>&</sup>lt;sup>4</sup> In the context of this guidance, sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.

# Appendix B. MAGIC GUIDELINES FOR STAGING AND GRADING ACUTE GVHD

## Acute GVHD Staging and Grading, MAGIC Guidelines

| Stage | Skin<br>(Active Erythema Only) | Liver<br>(Bilirubin) | Upper GI | Lower GI<br>(Stool Output/Day) |
|---|---|---|---|---|
| 0 | No active (erythematous)<br>GVHD rash | < 2 mg/dL | No or intermittent<br>nausea, vomiting, or<br>anorexia | Adult: < 500 mL/day or<br>< 3 episodes/day.<br>Child: < 10 mL/kg per day<br>or < 4 episodes/day. |
| 1 | Maculopapular rash<br>< 25% BSA | 2-3 mg/dL | Persistent nausea,<br>vomiting, or anorexia | Adult: 500-999 mL/day or 3-4 episodes/day. Child: 10-19.9 mL/kg per day or 4-6 episodes/day. |
| 2 | Maculopapular rash<br>25%-50% BSA | 3.1-6 mg/dL | - | Adult: 1000-1500mL/day or 5-7 episodes/day. Child: 20-30 mL/kg per day or 7-10 episodes/day. |
| 3 | Maculopapular rash<br>> 50% BSA | 6.1-15 mg/dL | - | Adult: > 1500 mL/day or<br>> 7 episodes/day.<br>Child: > 30 mL/kg per day<br>or > 10 episodes/day. |
| 4 | Generalized erythroderma<br>(>50%) with bullae | > 15 mg/dL | - | Severe abdominal pain with<br>or without ileus or grossly<br>bloody stool (regardless of<br>stool volume). |

Overall clinical grade (based on most severe target organ involvement):

Grade 0: No stage 1-4 of any organ.

Grade I: Stage 1-2 skin without liver, upper GI, or lower GI involvement.

Grade II: Stage 3 rash and/or stage 1 liver and/or stage 1 upper GI and/or stage 1 lower GI.

Grade III: Stage 2-3 liver and/or stage 2-3 lower GI, with stage 0-3 skin and/or stage 0-1 upper GI.

Grade IV: Stage 4 skin, liver, or lower GI involvement, with stage 0-1 upper GI.

#### **Response Definitions:**

GVHD response assessments will be made with respect to changes in the organ stage relative to Study Day 1.

- Complete response (CR) is defined as a score of 0 for the GVHD grading in all evaluable organs. For a response to be scored as CR at Day 28 or later, the participant must still be in CR on that day and have had no intervening additional therapy for an earlier progression, mixed response (MR), or no response (NR).
- Very good partial response (VGPR) is defined as follows:
  - Skin: No rash, or residual erythematous rash involving < 25% of the body surface, without bullae (residual faint erythema and hyperpigmentation do not count).
  - Liver: Total serum bilirubin concentration < 2 mg/dL or < 25% of baseline at enrollment.
  - Gut:
    - Tolerating food or enteral feeding.
    - o Predominantly formed stools.
    - o No overt gastrointestinal bleeding or abdominal cramping.
    - No more than occasional nausea or vomiting.
- Partial response (PR) is defined as improvement in 1 stage in 1 or more organs involved with GVHD symptoms without progression in others. For a response to be scored as PR at Day 28 or later, the participant must still be in PR on that day and have had no intervening additional therapy for an earlier progression, MR, or NR.
- Mixed response is defined as improvement in 1 or more organs with deterioration in another organ manifesting symptoms of GVHD or development of symptoms of GVHD in a new organ.
- Progression of disease is defined as deterioration in at least 1 organ without any improvement in others.
- No response is defined as absence of any improvement or progression as defined.
   Subjects receiving secondary therapy (including need to re-escalate steroid dose to greater than the Day 1 dose) will be classified as nonresponders.

Source: CIBMTR 2009, Martin et al 2009, Harris et al 2016.

# APPENDIX C. CYTOCHROME P450 AND P-GLYCOPROTEIN INHIBITORS AND CYTOCHROME P450 INDUCERS

University of Washington School of Pharmaceutics: Drug Interaction Database Program. 2002. http://www.druginteractioninfo.org. Accessed May 2015. Highlighted rows indicate recent additions to the lists at the time the database search was performed.

# In Vivo CYP3A Inhibitors

| Inhibitor | Therapeutic Class | Inhibitor dosing (oral) | Object <sup>1</sup> (oral, unless otherwise specified) | AUC <sub>ratio</sub> | PMID or NDA# | Published |
|---|---|---|---|---|---|---|
| | | Potent CYP3A Inhibitors (yielding substrate AUCr > 5) | | | | |
| indinavir /RIT | Protease Inhibitors | 800/100 mg BID (1 day) | alfentanil | 36.5 | 19225389 | 2009 Mar |
| tipranavir/RIT | Protease Inhibitors | 500/200 mg BID (2 days) | <u>midazolam</u> | 26.91 | 20147896 | 2010 Jun |
| ritonavir | Protease Inhibitors | 3 doses of 100 mg over 24 h | <u>midazolam</u> | 26.41 | 20002087 | 2009 Dec |
| cobicistat (GS-9350) | None | 200 mg QD (14 days) | <u>midazolam</u> | 19.03 | 20043009 | 2010 Mar |
| indinavir | Protease Inhibitors | 800 mg TID (7 days) | vardenafil | 16.25 | NDA # 021400 | 2003 Aug |
| ketoconazole | Antifungals | 400 mg QD (4 days) | <u>midazolam</u> | 15.9 | 8181191 | 1994 May |
| troleandomycin | Antibiotics | 500 mg single dose | <u>midazolam</u> | 14.8 | 15536460 | 2004 Dec |
| telaprevir | Antivirals | 750 mg TID (16 days) | <u>midazolam</u> | 13.5 | 22162542 | 2012 Oct |
| danoprevir / RIT | Antivirals | 200/100 mg QD (14 days) | <u>midazolam</u> | 13.42 | 23872824 | 2013 Nov |
| elvitegravir / RIT | Treatments of AIDS | 150/100 mg QD (10 days) | midazolam | 12.8 | NDA # 203100 | 2012 |
| saquinavir / RIT | Protease Inhibitors | 1000/100 mg BID (14 days) | <u>midazolam</u> | 12.48 | 19792991 | 2009 Oct |
| lopinavir / RIT | Protease Inhibitors | 400/100 mg BID (2 days) | alfentanil | 11.47 | 24067429 | 2013 Dec |
| itraconazole | Antifungals | 200 mg QD (4 days) | midazolam | 10.8 | 8181191 | 1994 May |
| voriconazole | Antifungals | 200 mg BID (9 days) | midazolam | 9.63 | 21937987 | 2011 Nov |
| mibefradil | Calcium Channel Blockers | 100 mg single dose | midazolam | 8.86 | 14517191 | 2003 Oct |
| LCL161 | Cancer Treatments | 600 mg single dose | midazolam | 8.8 | 23585187 | 2013 Jun |
| clarithromycin | Antibiotics | 500 mg BID (7 days) | midazolam | 8.39 | 16432272 | 2006 Feb |
| posaconazole | Antifungals | 400 mg BID (7 days) | midazolam | 6.23 | 19302901 | 2009 Feb |
| telithromycin | Antibiotics | 800 mg QD (6 days) | midazolam | 6.2 | NDA# 021144 | 2004 |
| grapefruit juice DS <sup>2</sup> | Food Products | 240 mL TID (2 days) and 90 min, 60 min, 30 min prior to midazolam | midazolam | 5.95 | 12953340 | 2003 Aug |
| conivaptan | Diuretics | 40 mg BID (5 days) | midazolam | 5.76 | NDA # 021697 | 2005 |
| nefazodone | Antidepressants | 100-200 mg BID (12 days) | midazolam | 5.44 | 14551182 | 2003 Nov |
| nelfinavir | Protease Inhibitors | 1250 mg BID (14 days) | midazolam | 5.29 | 21406602 | 2011 Jun |
| saquinavir | Protease Inhibitors | 1200 mg TID (5 days) | midazolam | 5.18 | 10430107 | 1999 Jul |
| idelalisib | Kinase Inhibitors | 150 mg BID (8 days) | midazolam | 5.15 | NDA # 206545 | 2014 |
| boceprevir | Antivirals | 800 mg TID (6 days) | midazolam | 5.05 | NDA # 202258 | 2011 |
| | | Moderate CYP3A Inhibitors (AUCr ≥ 2 and < 5) | | | | |
| erythromycin | Antibiotics | 1000 mg single dose | midazolam | 4.99 | 25139487 | 2014 Dec |
| fluconazole | Antifungals | 400 mg single dose | midazolam | 4.93 | 16172184 | 2005 Oct |
| atazanavir / RIT | Protease Inhibitors | 300/100 mg BID | maraviroc | 4.9 | 18333863 | 2008 Apr |
| darunavir | Protease Inhibitors | 1200 mg BID (14 days) | saquinavir | 4.9 | NDA # 021976 | 2006 |
| diltiazem | Calcium Channel Blockers | 60 mg TID (2 days) | midazolam | 4.06 | 21209240 | 2011 Nov |
| darunavir / RIT | Protease Inhibitors | 400/100 mg BID (8 days) | sildenafil | 4.0 | NDA # 021976 | 2006 |
| dronedarone | Antiarrhythmics | 400 mg BID (14 days) | simvastatin | 3.66 | NDA # 022425 | 2009 |
| crizotinib | Kinase Inhibitors | 250 mg BID (28 days) | midazolam | 3.65 | NDA # 202570 | 2011 |
| atazanavir | Protease Inhibitors | 400 mg QD (7 days) | maraviroc | 3.57 | 18333863 | 2008 Apr |
| aprepitant | Antiemetics | 80-125 mg QD (5 days) | midazolam | 3.29 | 12891225 | 2003 Aug |
| casopitant | Antiemetics | 120 mg QD (14 days) | midazolam | 3.13 | 20840445 | 2010 Oct |
| amprenavir | Protease Inhibitors | 1200 mg BID (10 days) | rifabutin | 2.93 | 11158747 | 2001 Feb |
| imatinib | Antineoplastic Agents | 400 mg QD (7 days) | simvastatin | 2.92 | 14612892 | 2001 Peb |
| verapamil | Calcium Channel Blockers | 80 mg TID (2 days) | midazolam | 2.92 | 8198928 | 1994 Mar |
| | Antivirals | 30 mg QD (10 days) | | 2.69 | NDA # 205123 | 2013 |
| netupitant | Antiemetics | 300 mg single dose | simeprevir<br>midazolam | 2.44 | 23729226 | 2013 Oct |
| grapefruit juice | Food Products | 240 mL QD (4 days) | midazolam | 2.39 | 10546919 | 1999 Oct |
| <u> </u> | | | | 2.39 | | 2008 Jan |
| tofisopam | Benzodiazepines | 100 mg TID (9 days) | midazolam | | 17989974 | |
| cyclosporine | Immunosuppressants | Not provided (1-5 years) | midazolam<br>midazolam | 2.21 | 21753749 | 2011 Sep |
| ACT-178882 | Renin Inhibitors | 300 mg QD (14 days) | midazolam | | 22849770 | 2013 Dec |
| ciprofloxacin | Antibiotics | 500 mg single dose | sildenafil | 2.12 | 16372380 | 2005 Dec |
| schisandra sphenanthera | Herbal Medications | 3 capsules (= 11.25 mg deoxyschizandrin) BID (7 days) | midazolam | 2.05 | 19552749 | 2009 May |

| cimetidine | H-2 Receptor Antagonists | 200-400 mg QID (1.5 days) | midazolam | 2.02 | 6152615 | 1984 Sep |
|---|---|---|---|---|---|---|
| FK1706 | Central Nervous System Agents | 60 mg QD (14 days) | <u>midazolam</u> | 2.01 | 19889885 | 2010 Feb |
| lomitapide | Other Antilipemics | 60 mg QD (7 days) | simvastatin | 2.0 | NDA # 203858 | 2012 |
| | | Weak CYP3A Inhibitors (AUCr ≥ 1.25 and < 2) | | | | |
| tabimorelin | Hormone Replacement | 2.86-3.21 mg QD (7 days) | midazolam | 1.93 | 12610745 | 2003 Feb |
| ranolazine | Cardiovascular Drugs | 1000 mg BID (7 days) | simvastatin | 1.89 | NDA # 021526 | 2006 |
| amlodipine | Calcium Channel Blockers | 10 mg QD (9 days) | simvastatin | 1.8 | 23965645 | 2014 Apr |
| lomitapide | Other Antilipemics | 60 mg QD (7 days) | simvastatin | 1.77 | 24734312 | 2014 Mar |
| fosaprepitant (IV) | Antiemetics | 150 mg single 30-min infusion | midazolam | 1.76 | 21209230 | 2011 Dec |
| Seville orange juice | Food Products | 240 mL single dose | felodipine | 1.76 | 11180034 | 2001 Jan |
| amiodarone | Antiarrhythmics | 400 mg QD (4 days) | simvastatin acid | 1.76 | 17301736 | 2007 May |
| chlorzoxazone | Muscle Relaxants | 250 mg single dose (part of a 6-drug cocktail) | midazolam | 1.68 | 11736864 | 2001 Nov |
| M100240 | Antihypertensive Agents | 50 mg single dose | midazolam | 1.66 | 15051745 | 2004 Apr |
| fluvoxamine | Antidepressants | 50-00 mg BID (12 days) | midazolam | 1.66 | 14551182 | 2003 Nov |
| ranitidine | H-2 Receptor Antagonists | 150 mg BID (1.5 days) | midazolam | 1.66 | 6135440 | 1983 Jun |
| goldenseal | Herbal Medications | 1,323 mg (= 24.1 mg isoquinoline alkaloids) TID (14 days) | midazolam | 1.63 | 17495878 | 2008 Jan |
| clotrimazole | Antifungals | 10 mg TID (5 days) | midazolam | 1.61 | 20233179 | 2010 Feb |
| tacrolimus | Immunosuppressants | Not provided (1-5 years) | midazolam | 1.61 | 21753749 | 2011 Sep |
| cilostazol | Antiplatelets | 100 mg BID (7 days) | lovastatin | 1.56 | 10702889 | 1999 |
| ticagrelor | Antiplatelets | 180 mg bid (7 days) | simvastatin | 1.56 | NDA # 022433 | 2011 |
| peppermint oil | Food Products | 600 mg (= 300 uL peppermint oil) single dose | felodipine | 1.55 | 12235445 | 2002 Sep |
| ivacaftor | Cystic fibrosis treatments | 150 mg BID (6 days) | midazolam | 1.54 | NDA # 203188 | 2012 |
| GSK2248761 | Transcriptase Inhibitors | 100 mg QD (12 days) | midazolam | 1.54 | 22288567 | 2012 Aug |
| roxithromycin | Antibiotics | 300 mg QD (6 days) | midazolam | 1.47 | 7995324 | 1994 |
| suvorexant | Hypnotics - Sedatives | 80 mg QD (14 days) | midazolam | 1.47 | NDA # 204569 | 2014 |
| propiverine | Anticholinergics | 15 mg BID (7 days) | midazolam | 1.46 | 16183781 | 2005 Dec |
| isoniazid | Antibiotics | 90 mg BID (4 days) | triazolam | 1.46 | 6140941 | 1983 Dec |
| berberine | Herbal Medications | 300 mg TID (14 days) | midazolam | 1.45 | 21870106 | 2012 Feb |
| oral contraceptives | Oral contraceptives | OC with low doses of estrogen (< 35 ug ethinylestradiol) (> 3 months) | triazolam | 1.44 | 6149030 | 1984 Nov |
| delavirdine | NNRTIs | 400 mg TID (9 days) | indinavir | 1.44 | 9665503 | 1998 Jul |
| daclatasvir | Antivirals | 60 mg QD (7 days) | simeprevir | 1.44 | NDA # 205123 | 2013 |
| faldaprevir | Antivirals | 240 mg BID (8 days) | ethinyl estradiol | 1.44 | 25385099 | 2015 Jan |
| simeprevir | Protease Inhibitors | 150 mg QD (11 days) | midazolam | 1.43 | NDA # 205123 | 2013 |
| atorvastatin | HMG CoA Reductase Inhibitors (Statins) | 10-40 mg/day (chronic treatment) | midazolam IV | 1.41 | 12911366 | 2003 Sep |
| tolvaptan | Vasopressin Antagonists | 60 mg single dose | lovastatin | 1.41 | NDA # 022275 | 2009 |
| almorexant | Hypnotics - Sedatives | 200 mg QD (9 days) | midazolam | 1.37 | 22990330 | 2013 Mar |
| GSK1292263 | Other Antilipemics | 300 mg BID (9 days) | simvastatin | 1.36 | 23256625 | 2013 Jun |
| linagliptin | Dipeptidyl Peptidase 4 Inhibitors | 10 mg QD (6 days) | simvastatin | 1.34 | 20497745 | 2010 Jun |
| resveratrol | Food Products | 1 g QD (4 weeks) | buspirone | 1.33 | 20716633 | 2010 Sep |
| lacidipine | Calcium Channel Blockers | 4 mg QD (8 days) | simvastatin | 1.33 | 11259986 | 2001 Feb |
| cranberry juice | Food Products | 240 mL double strength juice, 1 glass q 15 min x 3 | midazolam | 1.33 | 19114462 | 2009 Mar |
| pazopanib | Kinase Inhibitors | 800 mg QD (17 days) | midazolam | 1.32 | 20881954 | 2010 Nov |
| everolimus | Immunosuppressants | 10 mg QD (5 days) | midazolam | 1.31 | 23426978 | 2013 Apr |
| blueberry juice | Food Products | two doses of 300 mL, separated by 16 hours | buspirone | 1.31 | 22943633 | 2013 Apr |
| nilotinib | Kinase Inhibitors | 600 mg single dose | midazolam | 1.3 | NDA # 022068 | 2013 Apr |
| AMD070 | Fusion Inhibitors | 200 mg BID (8 days) | midazolam | 1.29 | 18362694 | 2007<br>2008 Apr |
| alprazolam | Benzodiazepines | 1 mg TID (7 days) | buspirone | 1.29 | 8300893 | 1993 Nov |
| bicalutamide | Antiandrogens | 150 mg QD (>3 months) | midazolam | 1.27 | 15509184 | 2004 |
| sitaxentan | Endothelin Receptor Antagonists | 100 mg QD (7 days) | sildenafil | 1.27 | 20078609 | 2010 Jan |
| | | | | 1.27 | | |
| azithromycin | Antibiotics Herbal Medications | 500 mg QD (3 days) | midazolam | 1.25 | 8720318<br>17050793 | 1996 Feb<br>2006 Nov |
| ginkgo<br>teriflunomide | | 120 mg TID (28 days) | midazolam<br>midazolam | 1.25 | NDA # 202992 | 2006 Nov<br>2012 |
| | Other Immunomodulators | 14-70 mg QD (14 days) | <u>midazolam</u> | 1.25 | NUA # 202992 | 2012 |

<sup>&</sup>lt;sup>1</sup> To allow better comparability, DDI studies with the probe substrate midazolam were selected first.

When no study with midazolam was available, the AUCratio of another probe or sensitive substrate is presented.

<sup>&</sup>lt;sup>2</sup> 240 mL GFJ double-strength administered TID for 3 days

# In Vivo CYP3A Inducers

| Inducers | Therapeutic class | Object (oral, unless otherwise specified) | % ↓ AUC | % ↑ oral CL | Precipitant Dose (oral) | PMID or NDA# | Published |
|---|---|---|---|---|---|---|---|
| | Poter | | ed by ≥ 80% or ( | CL increased by | more than 5 fold (400%)) | | |
| rifampin | Antibiotics | budesonide | 99.7 | 36904.5 | 600 mg QD (7 days) | 15726657 | 2005 Mar |
| mitotane | Other Antineoplastics | midazolam | 94.5 | Not Provided | maximum of 3.5 g TID (chronic therapy) | 21220434 | 2011 Apr |
| avasimibe | Other Antilipemics | midazolam | 93.5 | Not Provided | 750 mg/day (7 days) | 12766253 | 2003 Sep |
| phenytoin | Anticonvulsants | nisoldipine | 89.5 | Not Provided | 200-450 mg/day (chronic treatment) | 8917062 | 1996 Nov |
| carbamazepine | Anticonvulsants | quetiapine | 86.6 | 643.1 | 200 mg TID (26 days) | 16390352 | 2006 Jan |
| enzalutamide | Antiandrogens | midazolam | 85.9 | Not Provided | 160 mg QD (85±3 days) | NDA # 203415 | 2012 |
| St John's Wort | Herbal Medications | midazolam | 80.0 | Not Provided | 300 mg TID (14 days) | 16341856 | 2006 Jan |
| rifabutin | Antibiotics | delavirdine | Not Provided | 458.0 | 300 mg QD (14 days) | 9224961 | 1997 Jun |
| phenobarbital | Anticonvulsants | verapamil | 76.6 | 400.9 | 100 mg QD (21 days) | 3392664 | 1988 Jul |
| | Mode | erate Inducers (AUC decr | eased by 50-809 | % or CL increase | d by 2-5 fold (100-400%)) | | |
| ritonavir and St. Johns wort | None | midazolam | 77.2 | Not Provided | ritonavir: 300 mg BID and SJW: 300 mg TID (14 days) | 19924124 | 2010 Feb |
| semagacestat | Alzheimer's Treatments | midazolam | 76.4 | 324.6 | 140 mg QD (10 days) | 22789530 | 2012 Oct |
| efavirenz | NNRTIs | alfentanil | 76 | 369.4 | 600 mg QD (20 days) | 22398970 | 2012 Apr |
| tipranavir and ritonavir | Protease Inhibitors | saquinavir | 75.6 | Not Provided | tipranavir: 500 mg and ritonavir: 200 mg BID (14 days) | 18176328 | 2008 Apr |
| bosentan | Endothelin Receptor Antagonists | sildenafil | 69.0 | 239.8 | 62.5-125 mg BID (8 weeks) | 15963102 | 2005 Jul |
| genistein | Food Products | midazolam | 13.7 | 136.9 | 1000 mg QD (14 days) | 21943317 | 2012 Feb |
| thioridazine | Antipsychotics | quetiapine | 68.7 | 104.5 | 100-300 mg QD (15 days) | 22569350 | 2012 Jun |
| nafcillin | Antibiotics | nifedipine | 62.6 | 145.1 | 500 mg 4 times daily (5 days) | 12814453 | 2003 Jun |
| talviraline | NNRTIs | indinavir | 61.7 | 181.2 | 500 mg TID (14 days) | 10516944 | 1999 Oct |
| lopinavir | Protease Inhibitors | amprenavir | 59.7 | Not Provided | 400 mg BID (4 weeks) | 15060509 | 2004 Apr |
| modafinil | Psychostimulants | triazolam | 57.6 | 35.7 | 200-400 mg QD (28 days) | 11823757 | 2002 Jan |
| etravirine | NNRTIs | sildenafil | 56.7 | Not Provided | 800 mg BID (13.5 days) | NDA# 022187 | 2008 |
| lersivirine | NNRTIs | midazolam | 51.4 | 105.5 | 1000 mg BID (14 days) | 22527351 | 2012 Nov |
| | Wea | k Inducers (AUC decrease | ed by 20-50% or | CL increased by | less than 2 fold (100%)) | | |
| eslicarbazepine | Anticonvulsants | simvastatin | 49.4 | 98.4 | 800 mg QD (14 days) | 23726291 | 2013 Sep |
| telaprevir | Antivirals | darunavir | 48.4 | Not Provided | 1125 mg BID (4 days) | NDA# 201917 | 2011 |
| garlic | Food Products | saquinavir | 44.7 | Not Provided | caplet of GarliPure BID (20 days) | 11740713 | 2002 Jan |
| bexarotene | Other Antineoplastics | atorvastatin | 45.3 | Not Provided | 400 mg/m2 QD (at least two 4-week cycles) | 22057855 | 2012 Feb |
| amprenavir | Protease Inhibitors | lopinavir | 43.0 | Not Provided | 700 mg BID (2-4 weeks) | 15668539 | 2005 Jan |
| raltegravir | HIV-Integrase Strand Transfer Inhibitors | darunavir | 42.0 | Not Provided | 400 mg BID | 21958880 | 2012 Feb |
| vemurafenib | Kinase Inhibitors | midazolam | 39.4 | Not Provided | 960 mg BID (15 days) | NDA # 202429 | 2011 |
| troglitazone | Thiazolidinediones | simvastatin | 37.7 | Not Provided | 400 mg QD (24 days) | 11361054 | 2001 May |
| sorafenib | Kinase Inhibitors | sirolimus | 36.9 | Not Provided | 200 mg BID (11 days) | 21045832 | 2010 Nov |
| rufinamide | Anticonvulsants | triazolam | 36.7 | 53.4 | 400 mg BID (11.5 days) | NDA # 021911 | 2008 |
| pleconaril | Antivirals | midazolam | 34.6 | 52.8 | 400 mg TID (6 days) | 16467135 | 2006 May |
| ginseng | Herbal Medications | midazolam | 34.2 | 50.7 | 500 mg BID (28 days) | 21646440 | 2012 Jun |
| boceprevir | Antivirals | darunavir | 34.2 | 41.0 | 800 mg every 8 hrs (6 days) | 23155151 | 2013 Mar |
| sulfinpyrazone | Antigout and Uricosuric Agents | cyclosporine | 33.9 (cha | inge in C <sub>avg</sub> ) | 200 mg/day | 11124491 | 2000 Dec |
| gingko | Herbal Medications | midazolam | 33.7 | 52.6 | 120 mg BID (28 days) | 18205997 | 2008 Feb |
| vinblastine | Vinca Alkaloids | midazolam IV | 33.2 | 48.8 | not provided (4 cycles) | 20959500 | 2010 Nov |
| nevirapine | NNRTIs | indinavir | 32.5 | Not Provided | 200 mg QD (14 days), then BID (19 days) | 10191212 | 1999 May |
| armodafinil (R-modafinil) | Psychostimulants | midazolam | 32.2 | 54.7 | 100-250 mg/day (31 days) | 18076219 | 2008 |
| ticagrelor | Anticoagulants and Antiplatelets | midazolam | 31.7 | 46.5 | 400 mg QD (6 days) | 23870610 | 2013 Jul |
| LCL161 | Cancer Treatments | midazolam | 29.8 | 34.0 | 600 mg single dose | 23585187 | 2013 Jun |
| vicriviroc and ritonavir | Treatments of AIDS | ethinyl estradiol | 29.4 | Not Provided | 30 mg vicriviroc and 100 mg ritonavir QD (10 days) | 22015327 | 2011 Oct |

#### Incyte Corporation Protocol INCB 18424-271 Amendment 2

| ritonavir | Protease Inhibitors | ethinyl estradiol | 29.2 | Not Provided | 100 mg QD (10 days) | 22015327 | 2011 Oct |
|---|---|---|---|---|---|---|---|
| prednisone | Corticosteroids | tacrolimus | 29.0 | Not Provided | 1.5 mg/kg/day | 15787787 | 2005 Apr |
| oxcarbazepine | Anticonvulsants | felodipine | 28.1 | Not Provided | 450 mg BID (7 days) | 8451779 | 1993 Feb |
| danshen | Herbal Medications | midazolam | 27.9 | 32.8 | 4 g TID (14 days) | 20565457 | 2010 Jun |
| clobazam | Benzodiazepines | midazolam | 27.7 | Not Provided | 40 mg QD (15 days) | 22422635 | 2012 Apr |
| echinacea | Herbal Medications | midazolam | 27.3 | 37.5 | 500 mg TID (28 days) | 20393696 | 2010 Aug |
| ticlopidine | Anticoagulants and Antiplatelets | alfentanil | 27.0 | 50.0 | 250 mg BID (4 days) | 23361846 | 2013 Mar |
| brivaracetam | Anticonvulsants | ethinyl estradiol | 26.8 | 37.3 | 200 mg BID (21 days) | 24386664 | 2013 Dec |
| Stribild* | Treatments of AIDS | ethinyl estradiol | 26.2 | 31.3 | 150 mg ELV + 150 mg COB + 200 mg EMT+ 300 mg TEN | NDA # 203100 | 2012 |
| pioglitazone | Thiazolidinediones | midazolam | 26.0 | Not Provided | 45 mg QD 7 days | Actos® Product Label | |
| dexamethasone | Corticosteroids | aprepitant | 25.0 | Not Provided | 8 mg/day (5 days) | NDA # 021549 | 2003 |
| terbinafine | Antifungals | midazolam | 24.5 | Not Provided | 250 mg QD (4 days) | 8527290 | 1995 Sep |
| quercetin | Food Products | midazolam | 23.6 | Not Provided | 500 mg QD (13 days) | 21680781 | 2012 Jun |
| glycyrrhizin | Herbal Medications | midazolam | 23.0 | Not Provided | 150 mg BID (15 days) | 20393696 | 2010 Aug |
| aprepitant | Neurokinin-1 Receptor Antagonists | midazolam IV | 22.1 | 28.5 | 125/80 mg QD (3 days) | 14973304 | 2004 Mar |
| PA-824 | Antibiotics | midazolam | 22.1 | 20.7 | 400 mg QD (14 days) | 23689718 | 2013 Aug |
| oritavancin | Antibiotics | midazolam | 18.7 | 23.9 | 1200 mg IV single infusion | NDA # 206334 | 2014 |
| AZD 7325 | Anxiolytics | midazolam | 18.7 | 22.6 | 10 mg QD (12 days) | 22122233 | 2012 Jul |
| methylprednisolone | Corticosteroids | cyclosporine | 15.8 | 35.0 | 16 mg/day (12 days) then 8 mg/day (6 months) | 12164891 | 2002 Sep |
| topiramate | Anticonvulsants | ethinyl estradiol | 12.0 | 20.2 | 50 mg/day (21 days) | 12681003 | 2003 Apr |

<sup>1-</sup> Ritonavir has dual effects of simultaneous CYP3A inhibition and induction, and the net pharmacokinetic outcome during chronic ritonavir therapy is inhibition of CYP3A activity.

<sup>2-</sup> All the substrates presented in the table are sensitive CYP3A substrates (see definition in FDA guidance) except verapamil, cyclosporine, ethinyl estradiol, and delavirdine.

<sup>\*</sup> Stribild is a combination of elvitegravir, cobicistat, emtricitabine and tenofovir DF

Signature Manifest Page 1 of 1

## Signature Manifest

Document Number: IC-DEV-PROT-AMEND-0191

Title: INCB 18424-271 Protocol Amendment 2

Revision: 0

All dates and times are in Eastern Standard Time.

#### APPROVAL: 18424-271 Amendment 2

#### Rejection Collaboration Title Name/Signature Date Meaning/Reason 06 Oct 2016, 10:19:23 AM Complete **Approval and Release** Title Meaning/Reason Name/Signature Date 06 Oct 2016, 10:21:45 AM Approved 06 Oct 2016, 10:35:19 AM Approved 06 Oct 2016, 10:42:11 AM Approved 06 Oct 2016, 11:48:55 AM Approved